

# NCT #NCT03564145

# Statistical Analysis Plan

Sol-Gel Technologies Ltd. SGT-54-07

Version: 1.0 Date: 18 NOV 2019

# STATISTICAL ANALYSIS PLAN

Protocol Number: SGT-54-07

Study Title: A Multi-Center, Open-Label, Long-Term

Safety Study of S5G4T-1 to Evaluate the Safety of S5G4T-1 in Papulopustular

Rosacea Patients

Development Phase of Study: 3

Sponsor: Sol-Gel Technologies Ltd.

Sponsor Contact:

Statistical Analysis Plan based on Protocol Version: 4.0

Statistical Analysis Plan Date: 18NOV2019

Statistical Analysis Plan Version: V1.0



Sol-Gel Technologies Ltd. SGT-54-07 Version: 1.0

Date: 18 NOV 2019

SAP Approval

Authored by:

| | _ | | |
|---------------------------|----|-------|-------------|
| SIGNATURE: | | DATE: | 19Nov 2019 |
| QST Consultations, Ltd. | | | |
| Reviewed by: | | | |
| SIGNATURE: | | DATE: | 19 NOV 2019 |
| QST Consultations, Ltd. | | | |
| Approved by: | | | |
| SIGNATURE: | | DATE: | |
| | -1 | _ | |
| Sol-Gel Technologies Ltd. | | | |

Revisions to the Statistical Analysis Plan described herein must be approved through a formal written amendment with the exception of minor editorial changes to tables, figures, or listing shells, and any necessary textual clarifications for programmers that do not affect the stated analysis variables, study endpoints, or statistical methods.




# SAP Change History

| Version | Date | Summary of Changes | Author |
|---------|-----------|--------------------|--------|
| 1 | 18NOV2019 | Original document | |




# **TABLE OF CONTENTS**

| 1. | LIS | T OF A | BBREVIATIONS AND DEFINITIONS OF TERMS | 6 |
|---|---|---|---|---|
| 2. | PRI | EFACE | | 7 |
| 3. | RES | SPONSI | BILITIES | 7 |
| | | | CTION | |
| 4. | 1111 | KUDU | CHON | |
| <b>5.</b> | STU | JDY OB | BJECTIVES | 9 |
| 6. | STU | J <b>DY DE</b> | SIGN | 10 |
| | 6.1 | | l Study Design | |
| | | 6.1.1 | Schedule of Visits and Assessments | 11 |
| | | 6.1.2 | Method of Assigning Subjects to Treatment Groups | 11 |
| | | 6.1.3 | Blinding | |
| 7. | FFI | TICACY | AND SAFETY ENDPOINTS | 12 |
| /• | 7.1 | | ey Endpoints | |
| | 7.2 | | Endpoints | |
| | | _ | | |
| 8. | | | CAL AND ANALYTICAL PLANS | |
| | 8.1 | | ıl Methodology | |
| | | 8.1.1 | Statistical Analysis | |
| | | 8.1.2 | Baseline Definition | |
| | | 8.1.3 | Visit Windowing | |
| | | 8.1.4 | Adjustments for Covariates | |
| | | 8.1.5 | Handling of Dropouts or Missing Data | |
| | | 8.1.6 | Interim Analyses and Data Monitoring | |
| | | 8.1.7 | Multicenter Studies | 17 |
| | | 8.1.8 | Multiple Comparisons/Multiplicity | 17 |
| | | 8.1.9 | Use of an Efficacy Subset of Subjects | 17 |
| | | 8.1.10 | Active-Control Studies Intended to Show Equivalence | 17 |
| | | 8.1.11 | Examination of Subgroups | 17 |
| | 8.2 | Dispos | ition of Subjects | 17 |
| | 8.3 | Protoco | ol Deviations | 18 |
| | 8.4 | Data S | ets Analyzed | 18 |
| | | 8.4.1 | Safety Population | 18 |




| | 8.5 | Demog | graphic and | Other Baseline Characteristics | 18 |
|---|---|---|---|---|---|
| | 8.6 | Prior a | nd Concom | nitant Medications | 19 |
| | 8.7 | Prior a | nd Concom | nitant Procedures/Therapies | 19 |
| | 8.8 | Analys | sis of Effica | acy | 20 |
| | | 8.8.1 | IGA | | 20 |
| | | 8.8.2 | Retreatme | ents | 20 |
| | | | 8.8.2.1 | RosaQoL21 | |
| | | | 8.8.2.2 | Rosacea Erythema and Telangiectasia Assessments | 22 |
| | 8.9 | Safety | Evaluation | | |
| | | 8.9.1 | Extent of | Exposure | 22 |
| | | 8.9.2 | Adverse 1 | Events | 23 |
| | | 8.9.3 | | Laboratory Evaluation | |
| | | 8.9.4 | Other Ob | servations Related to Safety | 24 |
| | | | 8.9.4.1 | Cutaneous Safety Assessments | 24 |
| | | | 8.9.4.2 | Local Tolerability Assessments | |
| | | | 8.9.4.3 | Vital Signs | |
| | | | 8.9.4.4 | Physical Examination | 25 |
| 9. | <b>DE</b> | ΓERMI | NATION ( | OF SAMPLE SIZE | 25 |
| 10. | СН | ANGES | S IN THE I | PLANNED ANALYSES | 25 |
| 11. | REI | FEREN | CES | | 25 |
| 12. | INI | DEX OF | PLANNE | D TABLES | 27 |
| 13. | INI | DEX OF | PLANNE | D LISTINGS | 96 |



Sol-Gel Technologies Ltd. SGT-54-07

Version: 1.0

Date: 18 NOV 2019

#### 1. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE(s) adverse event(s)

ATC Anatomical Therapeutic Chemical

BMI body mass index BPO benzoyl peroxide

C Celsius

cm centimeters

CRF(s) case report form(s)
CI confidence interval

eCRF(s) electronic case report form(s)
E-BPO encapsulated benzoyl peroxide

ET early termination

IGA Investigator Global Assessment
IWRS Interactive Web Response System

kg kilograms
max maximum
min minimum

n number of observations

N number of subjects (sample size)

PI Principal Investigator
QST QST Consultations, Ltd.

RosaQoL Rosacea Quality of Life Questionnaire

SAE(s) serious adverse event(s) SAP Statistical Analysis Plan

SAS® Statistical Analysis System (SAS® Institute Inc., Cary, NC)

SD standard deviation SOC system organ class

TEAE(s) treatment-emergent adverse event(s)

WHO World Health Organization



Sol-Gel Technologies Ltd. SGT-54-07


#### 2. PREFACE

This Statistical Analysis Plan (SAP) describes the statistical analyses as it is foreseen before the database is locked. The SAP will serve as a compliment to the study protocol and supersedes it in case of differences. In case of major differences between the study protocol and SAP, e.g. changes in the analysis related to the primary endpoint, a protocol amendment will be considered. The SAP may be updated during the study conduct and will be finalized before the database lock.

The following documents were reviewed in preparation of this SAP:

- Clinical Study Protocol SGT-54-07
  - o Version 1.0 issued on 27JUN2018,
  - o Version 2.0 issued on 20AUG2018,
  - o Version 3.0 issued on 16SEP2018,
  - Version 4.0 issued on 27NOV2018
- Case report form (CRF) for SGT-54-07.
- ICH E9 Guidance on Statistical Principles for Clinical Trials.
- ICH E3 Structure and Content of Clinical Study Reports (CSRs)

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a patient in this study.

#### 3. RESPONSIBILITIES

The study statistician will be responsible for the statistical analysis planning. QST Consultations, Ltd. (QST), a Contract Research Organization selected by Sol-Gel, will be responsible for the execution of all statistical programming deliverables. The statistical programming work will be supervised by the study statistician.

#### 4. INTRODUCTION

S5G4T-1 is an innovative topical formulation containing 5% encapsulated benzoyl peroxide (E-BPO) that Sol-Gel is developing for the treatment of rosacea. If approved, S5G4T-1 will be the




Date: 18 NOV 2019

first product containing E-BPO for the treatment of rosacea. Sol-Gel believes S5G4T-1 has the potential to be as tolerable as, and more effective than, currently marketed rosacea drugs.

Rosacea is a chronic and recurrent inflammatory dermatological disorder of unknown etiology. The disease is common, especially in fair-skinned people of Celtic and northern European heritage. The onset of the disorder is usually between the ages of 30 and 50. Early stages of the disease affect women more often than men at a ratio of 3 to 1 [3, 5]. Rosacea usually starts as flushing and subtle redness on the cheeks, nose, chin or forehead. Alcohol, hot drinks, spicy foods, stress, sunlight and extreme heat or cold can trigger the onset of this disease. If left untreated, rosacea can slowly worsen over time. As the condition progresses, patients experience inflammatory lesions (papules and pustules), vivid erythema and telangiectasia. Patients may develop furuncles, cystic nodules, granulomas and tissue hypertrophy, sometimes leading to rhinophyma.

The first report on the treatment of rosacea with benzoyl peroxide (BPO) as a single agent was described by in Montes *et al.* in 1983 [6]. In this limited study, 5% BPO, after 5 to 8 weeks of treatment, demonstrated superiority compared to control with respect to papules, pustules and erythema but not telangiectasia. The formulation was a basic formulation with BPO dissolved and delivered in acetone. Irritation and burning was reported in both groups, most likely due to the well-known effects of BPO.

More recently, Breneman *et al.* 2004 [1] published the results of a study in collaboration with J. Leyden. This study was a double-blind, vehicle-controlled study, using a combination gel product of 5% BPO and 1% clindamycin to treat patients having moderate to severe rosacea. The most dramatic effect of the BPO/clindamycin treatment was on the reduction of papules and pustules. Side effects included the well-known effects of BPO, burning and itching.

The most prevalent AEs associated with topical BPO were related to local irritation. These included dry skin, peeling, burning and erythema. For the published studies, the percentage of subjects with dermatological AEs considered possibly related to BPO monotherapy ranged from 7% [7] to 22% [8]. In studies sponsored by Sol-Gel, the percentage of subjects with dermatological AEs associated with E-BPO 7% cream ranged from 0% (Study SGT-03B) to 37% (Study SGT-04), and the incidence of dermatological AEs associated with lower concentrations of E-BPO cream was  $\leq 2\%$ .

Several published studies reported AEs that might be associated with sensitivity of subjects to BPO. Leyden *et al.* 2001 [4] reported that 1 of 164 subjects (0.6%) receiving 5% BPO had an allergic reaction, and that allergic reactions occurred for 1.2% of subjects receiving 5% BPO plus 1% clindamycin and for 3.1% of subjects receiving 5% BPO plus 3% erythromycin. Tschen *et* 




Date: 18 NOV 2019

al. 2001 [8] reported a rash for 1 of 95 subjects (1%) that received 5% BPO monotherapy. Fyrand and Jakobsen 1986 [2] reported that 2 of 49 subjects withdrew from the study due to severe dermatitis indicating possible sensitization. Montes et al. 1983 [6] reported hypersensitivity to BPO in 4 of 31 subjects receiving 5% BPO acetone gel for rosacea. Weiss et al. 2002 [9] reported that 2 of 257 subjects receiving BPO plus clindamycin developed urticaria. In Study KGL 5782, 1 subject developed possible delayed contact hypersensitivity to both E-BPO, 2.5%, and Proactiv, 2.5%, indicating the hypersensitivity was probably due to BPO not an excipient. None of these events that might possibly indicate sensitization were confirmed by patch testing.

In 2012, Sol-Gel completed a double blind, randomized, dose-ranging Phase 2 trial for S5G4T-1 involving 92 adult patients at 10 centers in the United States (Study SGT-EBPO1-09: A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Dose-Range Study of E-BPO Gel, 1% and 5%, and Vehicle Gel in the Treatment of Rosacea). The Phase 2 study had the primary endpoints: Success in Investigator Global Assessment (IGA) and reduction in the mean inflammatory lesion count at Week 12 (End of Study). Safety was evaluated through AE reporting and cutaneous safety and local tolerability assessments. Both E-BPO cream, 1% and 5% applied once daily for 12 weeks had a positive effect on rosacea and were safe and well tolerated in this study. No deaths or other SAEs were reported during the study. Study medication was withdrawn for 1 subject who applied E-BPO cream, 5% (severe application site reaction) and for 2 subjects who applied E-BPO cream, 1% (severe cyst and moderate application site dermatitis). None of the subjects had severe dryness, scaling, or pruritus post-baseline. One subject in the E-BPO cream, 5% group experienced severe stinging and burning reported as an AE.

#### 5. STUDY OBJECTIVES

The objective of this long-term safety study is to determine the nature, severity and frequency of the AE rate and the cutaneous safety and local tolerability assessments of S5G4T-1 when applied once daily, if applicable, for up to 52 weeks.

The safety endpoints to be assessed include the following:

- The frequency of both local and systemic AEs
- Investigator cutaneous safety assessment (dryness and scaling) and the local tolerability assessment (itching and burning/stinging) at Baseline and all post-baseline study visits.



Sol-Gel Technologies Ltd. SGT-54-07


#### 6. STUDY DESIGN

# 6.1 Overall Study Design

Approximately 700 patients will be enrolled at up to 56 sites. All patients in this open-label, long-term safety study will be assigned to treatment with S5G4T-1.

The objective of this study is to determine the long-term safety and tolerability of daily use of S5G4T-1 in papulopustular rosacea patients.

Patients who successfully completed the 12-week treatment period from Study SGT-54-01 or Study SGT-54-02 may be offered to continue in the long-term safety, open-label extension study (Study SGT-54-07) for up to an additional 40 weeks (sum of up to 52 weeks). The Sponsor may terminate the study once 300 patients complete a total of 28 weeks of treatment and 100 patients complete a total of 52 weeks.

Patients who completed the 12-week treatment period (± 4 days) for SGT-54-01 or SGT-54-02 and did not miss more than one visit (Visit 3, 4 or 5) in SGT-54-01 or SGT-54-02 will be admitted into the 54-07 study after the Entry Criteria have been met and an ICF has been signed. Qualified patients will receive study product at Baseline and will be treated for up to 40 weeks. At each visit, the patients will be assessed for a 5-point scale IGA of rosacea. If a patient is assessed as "clear" (0) or "almost clear" (1), the patient will not be dispensed the study product. If a patient is assessed as "mild", "moderate" or "severe" (score of 2, 3 or 4, respectively), study product will be dispensed and the patient will use the study product daily according to patient instructions. Rosacea Quality of Life Questionnaire (RosaQoL) will be completed at Baseline, Visits 5, 8, 11, and 14 and at End of Study or at early termination. The RosaQoL data of patients who were enrolled from SGT-54-01 or SGT-54-02, will be used from the questionnaire completed at Visit 6/Week 12 of SGT-54-01 or SGT-54-02. Rosacea erythema severity and telangiectasia assessments will be completed at all study visits. At each visit, the following safety measures will be recorded: monitoring for any local and systemic AEs, cutaneous safety (dryness, and scaling) and local tolerability (itching and burning/stinging) assessments on a scale ranging from 0 (None) to 3 (Severe), vital signs and physical examinations.

A urine pregnancy test is required at all visits for all females of child-bearing potential.

Clinical Evaluations will be performed at:

- 1. Visit 1/Screening, only applies for new patients
- 2. Visit 2/Baseline, Day 1 can also be Visit 6/Week 12, Day 85 of Study SGT-54-01 or Study SGT-54-02

TOOL.AN.10-01.01 Statistical Analysis Plan Template



Sol-Gel Technologies Ltd. SGT-54-07


- 3. Visit 3/Week 4, Day 29 (± 10 Days)
- 4. Visit 4/Week 8, Day 57 (± 10 Days)
- 5. Visit 5/Week 12, Day 85 (± 10 Days)
- 6. Visit 6/Week 16, Day 113 (± 10 Days)
- 7. Visit 7/Week 20, Day 141 (± 10 Days)
- 8. Visit 8/Week 24, Day 169 (± 10 Days)
- 9. Visit 9/Week 28, Day 197 (± 10 Days)
- 10. Visit 10/Week 32, Day 225 (± 10 Days)
- 11. Visit 11/Week 36, Day 253 (± 10 Days)
- 12. Visit 12/Week 40, Day 281 (± 10 Days)/ End of Treatment/End of Study for patients who complete the study, early terminate, or if the Sponsor terminates the study prematurely.

The study product will be administered in an open-label fashion, i.e., the treatment assignment will be known to the patient, to study personnel and Sol-Gel personnel and its representatives.

#### 6.1.1 Schedule of Visits and Assessments

The schedule of assessments can be found in Section 13.9 of the protocol.

# 6.1.2 Method of Assigning Subjects to Treatment Groups

All patients will receive S5G4T-1. The patient assignment schedule will be a stratified by investigational site. Patients will be assigned through the Interactive Web Response System (IWRS) a unique ID indicating pump number. The format of the supplied number of pump is XXXX. At each visit the patient will return the pump and will be dispensed the next pump according to the IWRS assignment.

# 6.1.3 Blinding

Not applicable.



Sol-Gel Technologies Ltd. SGT-54-07


#### 7. EFFICACY AND SAFETY ENDPOINTS

# 7.1 Efficacy Endpoints

This study is not intended to assess efficacy.

IGA is included to determine the need for treatment and subsequent re-treatment after treatment course (in either Study SGT-54-01 or Study SGT-54-02) and any subsequent 4-week courses, if applicable. Certain efficacy data and endpoints will, however, be summarized.

The number of retreatments and the number of treatment free days until the first retreatment (relapse) will be calculated as described in Section 8.7.2.2.

RosaQoL will be completed at Baseline, Visits 5, 8, 11, 14, and End of Study. The RosaQoL data of patients who were enrolled from SGT-54-01 or SGT-54-02, will be used from the questionnaire completed at Visit 6/Week 12 of SGT-54-01 or SGT-54-02.

Erythema severity and telangiectasia assessments will be completed at each study visit.

# 7.2 Safety Endpoints

Safety will be evaluated by monitoring AEs, and cutaneous safety (dryness and scaling) and local tolerability (itching and burning/stinging) assessments.

# 8. STATISTICAL AND ANALYTICAL PLANS

### 8.1 General Methodology

All statistical processing will be performed using SAS® version 9.4 or later unless otherwise stated.

Descriptive statistics will be used to provide an overview of the efficacy and safety results. For categorical parameters, the number and percentage of subjects in each category will be presented. For continuous parameters, descriptive statistics will include n (number of subjects), mean, standard deviation (SD), median, minimum (min) and maximum (max).

No inferential testing or imputations for missing data will be performed. No interim analyses are planned.

All analyses will be performed using the Safety Population of the study.

Where applicable the analysis will be presented by overall treatment group in 54-07 as well as by treatment group assignment in 54-01/54-02.

TOOL.AN.10-01.01 Statistical Analysis Plan Template



Sol-Gel Technologies Ltd. SGT-54-07


# 8.1.1 Statistical Analysis

All analyses will be performed by QST using SAS® Version 9.4 or later. All summary tables and data listings will be prepared utilizing SAS® software.

The standard operating procedures (SOPs) of QST will be followed in the creation and quality control of all data displays and analyses.

All data listings will be by subject. Additionally, all listings except the screen failure and randomization listings will be by treatment.

#### **8.1.2** Baseline Definition

Baseline is defined as the last non-missing assessment prior to first application in 54-01/02. For all subjects enrolled in 54-01/54-02, the baseline values from 54-01/54-02 will be considered the baseline values for calculations in 54-07. Missing results will not be flagged as baseline.

# 8.1.3 Visit Windowing

For subjects receiving S5G4T-1 in 54-01/54-02, data from 54-01/54-02 will be included in summaries of 54-07. For subjects receiving vehicle in 54-01/54-02, baseline values will be sourced from 54-01/54-02 and data from follow-up visits of 54-07 will be used in summaries. The table below details the analysis visits to be summarized and the associated visits from 54-01/54-02 or 54-07 which will be sourced for each type of subject.




Date: 18 NOV 2019

# **Analysis Visits for Efficacy and Safety Assessments**

| Analysis Visit | Subjects Receiving<br>S5G4T-1 in 54-01/54-02 | Subjects Receiving vehicle in 54-01/54-02 |
|---|---|---|
| Week 4 | 54-01/02 - Week 4 | 54-07 - Week 4 |
| Week 8 | 54-01/02 - Week 8 | 54-07 - Week 8 |
| Week 12 | 54-01/02 - Week 12 | 54-07 - Week 12 |
| Week 16 | 54-07 - Week 4 | 54-07 - Week 16 |
| Week 20 | 54-07 - Week 8 | 54-07 - Week 20 |
| Week 24 | 54-07 - Week 12 | 54-07 - Week 24 |
| Week 28 | 54-07 - Week 16 | 54-07 - Week 28 |
| Week 32 | 54-07 - Week 20 | 54-07 - Week 32 |
| Week 36 | 54-07 - Week 24 | 54-07 - Week 36 |
| Week 40 | 54-07 - Week 28 | 54-07 - Week 40 |
| Week 44 | 54-07 - Week 32 | Not available |
| Week 48 | 54-07 - Week 36 | Not available |
| Week 52 | 54-07 - Week 40 | Not available |

Data from 54-07 will be mapped to the appropriate analysis visit described above based on nominal visit indications. Data from Early Termination (ET) and unscheduled visits will be determined using analysis visit windows. The analysis visit windows for ET and unscheduled visits are presented in the following table.




Date: 18 NOV 2019

SGT-54-07 Analysis Visit Windows for Efficacy and Safety Assessments

| Nominal Visit | Target Study Day <sup>1</sup> | Window (Days) |
|---------------|-------------------------------|---------------|
| Week 4 | 29 | 22 to 42 |
| Week 8 | 57 | 43 to 70 |
| Week 12 | 85 | 71 to 98 |
| Week 16 | 113 | 99 to 126 |
| Week 20 | 141 | 127 to 154 |
| Week 24 | 169 | 155 to 182 |
| Week 28 | 197 | 183 to 210 |
| Week 32 | 225 | 211 to 238 |
| Week 36 | 253 | 239 to 266 |
| Week 40 | 281 | 267 to 294 |
| Week 44 | 309 | 295 to 322 |
| Week 48 | 337 | 323 to 350 |
| Week 52 | 365 | 351 to 378 |

<sup>&</sup>lt;sup>1</sup> Number of days since nominal Baseline visit of 54-07

Data collected at ET and unscheduled visits prior to study day 22 will not be analyzed. Data collected at ET and unscheduled visits after study day 378 will not be included in analyses.

The definition for the study day included in each study window is defined as below:

Study Day on or after Day 
$$1 = Visit Date - Day 1 Date + 1$$

If an assessment's mapped nominal visit is a visit at which the subject has data from a scheduled visit present, or if no analyses are planned for the assessment at the mapped nominal visit, the data collected at the ET or unscheduled visit will not be included in analyses.

In the event of multiple values from unscheduled or ET assessments within an analysis visit window, the value closest to the scheduled visit target study day will be used for analyses. If 2 values tie as closest to the time point (for example, one value is before and the other value is after the time point), then the later value will be selected.

Data collected at all visits will be included in the data listings with the 54-07 analysis visit presented.



Sol-Gel Technologies Ltd. SGT-54-07


# **8.1.4** Adjustments for Covariates

Not applicable to this study.

# 8.1.5 Handling of Dropouts or Missing Data

Incomplete start and end dates for medications will be imputed. Incomplete start dates for adverse events (AEs) will be imputed. Other data will not be imputed and will be summarized on an observed case basis.

# **8.1.5.1 Medication Date Imputation**

If the medication or procedure/therapy start date is incomplete, then it will be imputed as follows for the purpose of determining concomitant use:

- If the start date is completely missing, the start date will be equal to the first dose date. However, if the stop date is not missing and is before the first dose date, then the stop date will be used instead.
- If the start day is missing, the first day of the month will be used.
- If the start day and month are missing, then the first day of the first month (January) will be used.

If the medication or procedure/therapy stop date is incomplete, then it will be imputed as follows for the purpose of determining concomitant use:

- If the stop date is completely missing and the medication is not ongoing, the stop date will be equal to the last dose date or date of completion/withdrawal, whichever is the latest.
- If the stop day is missing, the last day of the month will be used.
- If the stop day and month are missing, then the last day of the last month (December) will be used.

# 8.1.5.2 Adverse Event Start Date Imputation

If the AE start date is incomplete, then it will be imputed as follows for the purpose of determining study day for the AE period breakdown described in Section 8.8.2:



Sol-Gel Technologies Ltd. SGT-54-07


- If the start date is completely missing, the start date will be equal to the first dose date. However, if the stop date is not missing and is before the first dose date, then the stop date will be used instead.
- If the start day is missing, the first day of the month will be used.
- If the start day and month are missing, then the first day of the first month (January) will be used.

# 8.1.6 Interim Analyses and Data Monitoring

No interim analysis or data monitoring is planned for this study.

#### **8.1.7** Multicenter Studies

The clinical study will be conducted under a common protocol for each investigational site with the intention of pooling all the data for analysis. Every effort will be made to promote consistency in study execution at each study site.

# 8.1.8 Multiple Comparisons/Multiplicity

No adjustments for multiple comparisons or multiplicity will be made.

# 8.1.9 Use of an Efficacy Subset of Subjects

Not applicable to this study.

# 8.1.10 Active-Control Studies Intended to Show Equivalence

Not applicable to this study.

# 8.1.11 Examination of Subgroups

Not applicable to this study.

#### 8.2 Disposition of Subjects

The number of subjects included in the Safety population will be summarized for all subjects, for subjects that received S5G4T-1 in 54-01/54-02, and for subjects that received vehicle in 54-01/54-02. The number of subjects enrolled, completed, and discontinued (including the reasons for discontinuation) will be summarized similarly.




Date: 18 NOV 2019

Subjects who are excluded from the Safety population will be summarized by the reasons for exclusion.

#### **8.3** Protocol Deviations

All protocol deviations will be reported to the sponsor and recorded throughout the study. Protocol deviations will not be entered into the database. SolGel will provide a list of protocol deviations to QST. A tabulation of protocol deviations will be presented in a data listing.

# 8.4 Data Sets Analyzed

Subjects will be presented/summarized based on the primary reason for exclusion.

# **8.4.1** Safety Population

All analyses will be performed using the Safety Population of the study. All patients who receive at least one confirmed dose of S5G4T-1 and have at least one assessment will be included in the Safety Population.

# 8.5 Demographic and Other Baseline Characteristics

All baseline summaries will be done on the Safety population.

Sex (categorical), race (categorical), and ethnicity (categorical) will be summarized by counts and percentages. Age (continuous), height (cm) (continuous), and weight (kilograms (kg)) (continuous), and body mass index (BMI) (continuous) will be summarized with descriptive statistics.

Age will be calculated as the difference in days between the date of birth and the date of informed consent and converted to years by dividing the number of days by 365.25 and using a floor function to drop the decimal portion. In case the exact birth day is missing, day 15 will be used. The BMI will be calculated as weight (kg) divided by squared height (m<sup>2</sup>).

Medical histories will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary and presented in a by-subject listing. All medical history for rollover subjects will be entered into 54-07 database and therefore medical history data will not be pulled from the 54-01 or 54-02 studies. The date of rosacea diagnosis for rollover subjects will be pulled from the 54-01 or 54-02 study.

The medical history data will be summarized with frequencies and percentages of patients with at least one medical history term reported, and patient frequencies and percentages on the System




Date: 18 NOV 2019

Organ Class (SOC) and Preferred Term levels. The number of events will also be summarized. The table will be sorted by overall descending frequency of SOC and then, within a SOC, by overall descending frequency of Preferred Term.

#### **8.6** Prior and Concomitant Medications

Concomitant medications will be coded to preferred name and Anatomical Therapeutic Chemical (ATC) classification of ingredients using the World Health Organization (WHO) Drug Global Dictionary, Format B3, Version March 1, 2018. Ongoing medications for rollover subjects will be entered into 54-07. Only medications that are not ongoing in 54-01 or 54-02 will be pulled forward for subjects who received S5G4T-1 in 54-01 or 54-02.

Medications which start prior to first application of S5G4T-1 (from 54-01/02 or 54-07) will be considered prior medications. Ongoing medications and medications ending after the date of first application (in 54-01/02 or 54-07) will be considered concomitant medications. If the date of first application is unknown and the medication is not listed as ongoing the interval will be considered "unknown". If the date of first application is unknown and the medication is listed as ongoing the interval will be considered concomitant.

Incomplete medication start and end dates will be imputed as described in Section 8.1.5.1.

A by-subject listing of all prior and concomitant medications will be presented for the Safety population.

#### 8.7 Prior and Concomitant Procedures/Therapies

Procedures/therapies will be coded using the MedDRA dictionary. Ongoing procedures/therapies for rollover subjects will be entered into 54-07. Only procedures/therapies that are not ongoing in 54-01 or 54-02 will be pulled forward for subjects who received S5G4T-1 in 54-01 or 54-02.

Procedures/therapies which start prior to first application of S5G4T-1 (from 54-01/02 or 54-07) will be considered prior procedures/therapies. Ongoing procedures/therapies and procedures/therapies ending after the date of first application (in 54-01/02 or 54-07) will be considered concomitant procedures/therapies. If the date of first application is unknown and the procedures/therapies is not listed as ongoing the interval will be considered "unknown". If the date of first application is unknown and the procedures/therapies is listed as ongoing the interval will be considered concomitant.

Incomplete procedures/therapies start and end dates will be imputed as described in Section 8.1.5.1.




Date: 18 NOV 2019

A by-subject listing of all prior and concomitant procedure/therapies will be presented for the Safety population.

### 8.8 Analysis of Efficacy

All efficacy analysis will be conducted on the Safety population.

#### 8.8.1 IGA

Descriptive statistics will be used to summarize the assessment of efficacy. IGA scores will be summarized at Baseline (see definition of baseline in Section 8.1.2) and every 4 weeks through end of the study. The number and percentage of patients who achieve treatment success at the scheduled study visits will be tabulated. A patient will be considered a success if their IGA score is clear or almost clear.

In addition to the above summary a by-subject listing of all IGA results will be presented.

#### 8.8.2 Retreatments

The number of retreatments is defined as the number of clinical confirmations of the condition for which the subject was initially treated after the first treatment period with S5G4T-1. For rollover subjects previously treated with vehicle, this is the number of treatments after the initial treatment in 54-07. For rollover subjects previously treated with S5G4T-1, this is the number of treatments in 54-07 following the cessation of the treatment which began in 54-01 or 54-02. A clinical confirmation of the condition will be defined as IGA no longer being clear or almost clear after a previous IGA of clear or almost clear. When a subject has a clear or almost clear IGA in 54-07, it is expected they were instructed not to dose until the IGA reached mild, moderate or severe.

The number of treatment free days until the first retreatment (relapse) will be calculated and summarized. Relapse will be defined as a subject no longer having an IGA of clear or almost clear after a previous visit IGA of clear or almost clear. When a subject has a clear or almost clear IGA in 54-07, it is expected they were instructed not to dose until the IGA reached mild, moderate or severe. Number of treatment free days until first retreatment is defined as the number of days between an initial IGA assessment of clear or almost clear while the subject was receiving S5G4T-1 until an IGA of mild, moderate or severe.

For rollover subjects previously treated with vehicle, the number of treatment free days will be the number of days between the end of their first treatment of S5G4T-1 in 54-07 (when the subject has an IGA of clear or almost clear) and the start of the next treatment in 54-07 (when the




Date: 18 NOV 2019

subject has an IGA indicating they should dose) if they treated with S5G4T-1 again or the end of the subject's participation in 54-07. For rollover subjects previously treated with S5G4T-1, the number of treatment free days will be the number of days between the end of the treatment that began in 54-01 or 54-02 (when the subject has an IGA of clear or almost clear) and the start of the next treatment in 54-07 (when the subject has an IGA indicating they should dose) if they treated with S5G4T-1 again or the end of the subject's participation in the 54-07.

Descriptive statistics for time to relapse (number of treatment free days until retreatment) and number of retreatments will be presented. A confidence interval (CI) for the median time to relapse will be presented using the Kaplan–Meier method. Patients who discontinue in 54-07 while not being treated and had not yet previously relapsed will be considered censored in the Kaplan–Meier analysis.

# 8.8.2.1 RosaQoL

The mean change in RosaQoL subscale scores from Baseline to Weeks 12, 24, 36, 48 and 52 will be summarized using descriptive statistics.

The subscores for the RosaQoL are computed as follows:

Total Score: the unweighted mean of all RosaQoL questions

Symptom subscale score: the unweighted mean of the following symptom questions

My rosacea burns or stings (item #2)

My rosacea is irritated (item #6)

My rosacea makes my skin sensitive (item #9)

My skin feels bumpy (uneven, not smooth, irregular) (item #16)

My skin flushes (item #17)

My skin gets irritated easily (cosmetics, aftershaves, cleansers) (item #18)

My eyes bother me (feels dry or gritty) (item #19)

Functional subscale score: the unweighted mean of the following functional questions

I try to cover up my rosacea (with make-up) (item #13)

I avoid certain foods or drinks because of my rosacea (item #15)

I avoid certain environments (heat, humidity, cold) because of my rosacea (item #21)

TOOL.AN.10-01.01 Statistical Analysis Plan Template




Sol-Gel Technologies Ltd. SGT-54-07


Emotion subscale score: the unweighted mean of the following emotion questions

I worry that my rosacea may be serious (item #1)

I worry about getting scars from my rosacea (item #3)

I worry that my rosacea may get worse (item #4)

I worry about side effects from rosacea medications (item #5)

I am embarrassed by my rosacea (item #7)

I am frustrated by my rosacea (item #8)

I am annoyed by my rosacea (item #10)

I am bothered by the appearance of my skin (redness, blotchiness) (item #11)

My rosacea makes me feel self-conscious (item #12)

I am bothered by persistence/reoccurrence of my rosacea (item #14)

I think about my rosacea (item #20)

Each individual item should be scored as follows: 1=Never, 2=Rarely, 3=Sometimes, 4=Often, and 5=All the time. Missing data values will not be used. If a subscale has items with missing results, the subscore and the total will not be calculated.

# 8.8.2.2 Rosacea Erythema and Telangiectasia Assessments

Rosacea erythema and telangiectasia assessments will be summarized at Baseline and every 4 weeks by counts and percentages. A by-subject listing will also be presented.

# 8.9 Safety Evaluation

# 8.9.1 Extent of Exposure

The extent of exposure to study product in each treatment group will be summarized by total number of days of exposure to S5G4T-1, total number of applications, number of missed applications, and number of applications the subject did not take because they were instructed not to dose. If the CRF reason for not dosing is anything but "Per Principal Investigator (PI) Instruction" it will be counted as a non-instructed missed dose. If the CRF reason for not dosing is "Per PI Instruction" it will be counted as an instructed missed dose.

The total number of days of exposure to S5G4T-1 is as follows:

TOOL.AN.10-01.01 Statistical Analysis Plan Template




Date: 18 NOV 2019

Date of last documented dose of S5G4T-1 - Date of first documented dose of S5G4T-1 +1

The total number of applications taken is as follows:

Sum of: [(End date of dosing interval from the CRF – Start date of dosing interval from the CRF + 1)\*Number of doses taking in dosing interval on CRF] for all dosing intervals on the CRF

The total number of non-instructed missed applications taken is as follows:

Sum of: (End date of dosing interval from the CRF with reason of "Other, specify reason" – Start date of dosing interval from the CRF + 1) for all dosing intervals on the CRF marked with a dose of 0 and with reason of "Other, specify reason".

The total number of instructed missed applications is as follows:

Sum of: (End date of dosing interval from the CRF with reason of "Per PI Instruction" – Start date of dosing interval from the CRF + 1) for all dosing intervals on the CRF marked with a dose of 0 and with reason of "Per PI Instruction".

Subjects who are lost to follow-up or have a dosing record with an unknown number of doses or unknown dates of the dosing intervals will not have extent of exposure variables calculated.

# **8.9.2** Adverse Events

AEs from 54-01/02 will be included in the analysis for 54-07. All AEs that were reported as ongoing in 54-01/02 will be added into the CRF for 54-07, while AEs reported as recovered/resolved will be pulled forward programmatically into 54-07.

AEs occurring during the study will be recorded and classified on the basis of MedDRA terminology. Descriptions of AEs will include the date of onset, the date the AE ended, the severity of the AE, the relationship to study product, the action taken regarding study product usage, the action taken to treat the AE, and the outcome. All reported treatment-emergent AEs (TEAEs) will be summarized by the number of patients reporting AEs, system organ class, severity, seriousness, and relationship to study product. TEAEs are those AEs with an onset on or after the date of the first study product application. For AEs recorded in the 54-07 study if the AE is not indicated as prior to first application on the CRF then it will be considered a TEAE. AEs from 54-01/02 for subjects who received S5G4T-1 in 54-01 or 54-02 will be considered a TEAE if they were considered at TEAE in the 54-01/02 study. AEs (including ongoing) from 54-01/02 study for subjects who received vehicle in 54-01 or 54-02 will be considered pre-treatment.




Date: 18 NOV 2019

AEs will be summarized by period (and total) and by severity. Each patient will be counted only once within a SOC or a Preferred Term by using the AEs with the highest severity within each category.

AEs will be summarized by period (and total) and by relationship to study product. Each patient will be counted only once within a system organ class or a preferred term by using the AEs with the greatest relationship within each category.

If relationship to study drug is reported as definitely, probably, or possible, then this is defined as related. If relationship to study drug is reported as unlikely or not related, then this is defined as unrelated.

TEAEs will be summarized in total as well as by the following periods based on time of onset in relation to date of first application of S5G4T-1, based on the definitions below. Start dates will be imputed as described in Section 8.1.5.2.

• 0-12 Weeks  $0 \le \text{onset day} \le 85$ 

• >12-28 Weeks  $86 \le \text{onset day} \le 197$ 

• >28-52 Weeks  $198 \le \text{onset day} \le 365$ 

• >52 Weeks onset day  $\geq$  366

All information pertaining to AEs noted during the study will be listed by patient, detailing verbatim given by the investigator, preferred term, system organ class, start date, stop date, severity, actions taken, and drug relatedness. The AE onset will also be shown relative (in number of days) to the day of initial application of the study product.

Serious adverse events (SAEs) will be tabulated by patient.

In addition, a list of patients who discontinued from the study and a list of patients who experienced SAEs will also be provided.

# 8.9.3 Clinical Laboratory Evaluation

Urine pregnancy test results will be presented in a by-subject listing.

# 8.9.4 Other Observations Related to Safety

# 8.9.4.1 Cutaneous Safety Assessments

Descriptive statistics by visit will be provided for dryness and scaling.

TOOL.AN.10-01.01 Statistical Analysis Plan Template



Sol-Gel Technologies Ltd. SGT-54-07


Cutaneous Safety Assessments will be presented in a by-subject listing.

# 8.9.4.2 Local Tolerability Assessments

Descriptive statistics by visit will be provided for itching and burning/stinging.

Local tolerability data will be presented in a by-subject listing.

# 8.9.4.3 Vital Signs

Vital sign measurements include heart rate (HR), sitting blood pressure (BP) (both systolic and diastolic), body temperature, and weight. The data will be summarized with descriptive statistics by visit. In addition, the changes from Baseline will be summarized with descriptive statistics.

Vital sign data will be presented in a by-subject listing.

# 8.9.4.4 Physical Examination

Physical examination data will be presented in a by-subject listing.

#### 9. DETERMINATION OF SAMPLE SIZE

The sample size for this study was based on the minimum requirement for a long-term safety study.

### 10. CHANGES IN THE PLANNED ANALYSES

The protocol was written in a way that subjects who did not participate in 54-01 or 54-02 could be enrolled into 54-07. When the SAP was created, 54-07 was fully enrolled, and no subject was enrolled who did not complete the 54-01 or 54-02 study. The SAP was written such that any text from the protocol that discusses the new subjects was excluded.

#### 11. REFERENCES

- 1. Breneman D, Savin R., VandePol C., Vamvakias G., Levy S., Leyden J. Double-blind, randomized, vehicle-controlled clinical trial of once-daily benzoyl peroxide/clindamycin topical gel in the treatment of patients with moderate to severe rosacea. *Int. J of Derm.* 2004; 43(5):381-387.
- 2. Fyrand O, Jakobsen HB. Water-based versus alcohol-based benzoyl peroxide preparations in the treatment of acne vulgaris. *Dermatolgica* 1986 172:263-267.



Sol-Gel Technologies Ltd. SGT-54-07


- 3. Jansen T and Plewig G. Rosacea: classification and treatment. JR Soc Med. 1997; 90(3):144-150.
- 4. Leyden JJ, Hickman JG, Jarratt MT, Stewart DM, Levy SF. The efficacy and safety of a combination benzoyl peroxide/clindamycin topical gel compared with benzoyl peroxide alone and a benzoyl peroxide/erythromycin combination product. *J Cutan Med Surg*. 2001. 5:37-42.
- 5. McDonnell JK and Tomecki KJ. Rosacea: an update. Clev Clinic J Med. 2000; 67(8):587-590.
- 6. Montes LF, Cordero AA., Kriner J., Loder J., Flanagan AD. Topical treatment of acne rosacea with benzoyl peroxide acetone gel. Cutis 1983; 32(2):185-190.
- 7. Thiboutot DM, Weiss J, Bucko A, Eichenfield L, Jones T, Clark S, Liu Y, Graeber M, Kang S. Adapalen-BPO Study Group. Adapalene-benzoyl peroxide, a fixed-dose combination for the treatment of acne vulgaris: results of a multicenter, randomized double-blind, controlled study. *J Am Acad Dermatol*. 2007. 57:791-799.
- 8. Tschen EH, Katz HI, Jones TM, Monroe EW, Kraus SJ, Connolly MA, Levy SF. A combination benzoyl peroxide and clindamycin topical gel compared with benzoyl peroxide, clindamycin phosphate, and vehicle in the treatment of acne vulgaris. *Cutis*. 2001. 67:165-169.
- 9. Weiss JW, Shavin J, Davis M. Preliminary results of a nonrandomized, multicenter, open-label study of patient satisfaction after treatment with combination benzoyl peroxide/clindamycin topical gel for mild to moderate acne. *Clin Ther*. 2002. 24:1706-1717.




# 12. INDEX OF PLANNED TABLES

| Table 14.0.1: Summary of Subject Completion/Discontinuation (All Enrolled Subjects)29 |
|---|
| Table 14.0.2.1: Summary of Subject Enrollment and Evaluability (All Enrolled Subjects)30 |
| Table 14.1.1.1: Summary of Subject Demographic Characteristics (Safety Population)31 |
| Table 14.1.2.1: Subject Baseline Characteristics (Safety Population)32 |
| Table 14.1.3.1: Summary of Medical History by System Organ Class and Preferred Term (Safety Population) |
| Table 14.1.4.1: Summary of Concomitant Medications by ATC Level 2 and Preferred Name (Safety Population) |
| Table 14.2.1.1: Summary of Investigator Global Assessment at Baseline and Week 40 (Safety Population) |
| Table 14.2.1.2: Summary of Investigator Global Assessment at Each Evaluation (Safety Population) |
| Table 14.2.2.1: Summary of RosaQoL Questionnaire Responses at Baseline and Week 40 (Safety Population) |
| Table 14.2.2.2: Summary of RosaQoL Questionnaire Responses at Each Evaluation (Safety Population) |
| Table 14.2.3: Summary of Erythema Assessment at Each Evaluation (Safety Population)54 |
| Table 14.2.4: Summary of Telangiectasia Assessment at Each Evaluation (Safety Population) 59 |
| Table 14.2.5: Summary of Reoccurrence (Safety Population) |
| Table 14.3.0.1: Summary of Extent of Exposure (Safety Population) |
| Table 14.3.1.1: Summary of Cutaneous Safety and Tolerability Evaluations (Safety Population) |
| Table 14.3.1.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population) |
| Table 14.3.1.2.2: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.2.3: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population) |
| Table 14.3.1.2.4: Summary of Treatment-Emergent Adverse Events by Relationship to Study Drug (Safety Population) |
| Table 14.3.1.3.1: Summary of Treatment-Emergent Adverse Event Characteristics - By Period (Safety Population) |




| Table 14.3.1.3.2: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term – By Period (Safety Population) |
|---|
| Table 14.3.1.3.3: Summary of Treatment-Emergent Adverse Events by Severity – By Period (Safety Population) |
| Table 14.3.1.3.4: Summary of Treatment-Emergent Adverse Events by Relationship to Study Drug – By Period (Safety Population) |
| Table 14.3.1.4.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population) |
| Table 14.3.1.4.2: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)84 |
| Table 14.3.1.4.3: Summary of Serious Treatment-Emergent Adverse Events by Severity (Safety Population)85 |
| Table 14.3.1.4.4: Summary of Treatment-Emergent Serious Adverse Events by Relationship to Study Drug (Safety Population) |
| Table 14.3.1.5.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics – By Period (Safety Population) |
| Table 14.3.1.5.2: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term – By Period (Safety Population) |
| Table 14.3.1.5.3: Summary of Treatment-Emergent Serious Adverse Events by Severity – By Period (Safety Population)90 |
| Table 14.3.1.5.4: Summary of Treatment-Emergent Serious Adverse Events by Relationship to Study Drug – By Period (Safety Population)91 |
| Table 14.3.1.4.1: Summary of Vital Signs (Safety Population)92 |



Table 14.0.1: Summary of Subject Completion/Discontinuation (All Enrolled Subjects)

| | SGT-54-01/SGT-54-02<br>Vehicle Cream | SGT-54-01/SG-54-02<br>E-BPO 5% Cream | SGT-54-07<br>E-BPO 5% Cream |
|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Completed Study | (IV MM) | (IV MIN) | (IV MM) |
| Yes | xx = (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Reason for Discontinuation | | | |
| Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost to Follow-Up | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lack of Efficacy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pregnancy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Protocol Violation | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Withdrawal by Subject | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Study Terminated by Sponsor | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Physician Decision | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Worsening of Condition | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.0.2.1: Summary of Subject Enrollment and Evaluability (All Enrolled Subjects)

| | SGT-54-01/SGT-54-02<br>Vehicle Cream<br>(N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| Number of Subjects Included in the Safety Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded from the Safety Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Reasons Excluded from the Safety Population <sup>a</sup> | | | |
| No Documented use of Study Drug | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No Post Baseline Safety Assessment | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Table includes primary reason (assigned in order presented in table) for reason subject was excluded.



Table 14.1.1.1: Summary of Subject Demographic Characteristics (Safety Population)

| | SGT-54-01/SGT-54-02 | SGT-54-01/SG-54-02 | SGT-54-07 |
|---|---|---|---|
| | Vehicle Cream | E-BPO 5% Cream | E-BPO 5% Cream |
| | (N=xxx) | N=xxx | (N=xxx) |
| Age (years) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Sex | | | |
| n | XX | XX | XX |
| Male | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Female | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Ethnicity | | | |
| n | XX | XX | XX |
| Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Reported/Unknown | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Race | | | |
| n | XX | XX | XX |
| American Indian or Alaska Native | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Asian | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Black or African American | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| White | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Multiple/Other <sup>a</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> See Listing 16.2.4.1 for a complete list of other races.

TOOL.AN.10-01.01 Statistical Analysis Plan Template




Table 14.1.2.1: Subject Baseline Characteristics (Safety Population)


| | SGT-54-01/SGT-54-02<br>Vehicle Cream<br>(N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| Height (cm) | (1. 1) | (2) | (11 11111) |
| n | XX | XX | xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Weight (kg) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| BMI (kg/m²) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |



Table 14.1.2.1: Subject Baseline Characteristics (Safety Population)


| | SGT-54-01/SGT-54-02<br>Vehicle Cream<br>(N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| Inflammatory Lesion Count | | · | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Investigator Global Assessment | | | |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Almost Clear | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 - Severe | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.1.3.1: Summary of Medical History by System Organ Class and Preferred Term (Safety Population)

| System Organ Class Preferred Term | E-BPO 5% Cream<br>(N=xxx) | |
|---|---|---|
| Number (%) of Subjects Reporting at Least One Medical History Term | By Subject <sup>a</sup> xx ( xx.x%) | By Event <sup>b</sup> |
| System Organ Class Preferred Term | xx ( xx.x%)<br>xx ( xx.x%) | xx<br>xx |

<sup>&</sup>lt;sup>a</sup> Counts reflect number of subjects reporting one or more medical history terms that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once. Percentages are based on the number of subjects in the safety population.

Note: MedDRA Version 21.0

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

{NOTE TO PROGRAMMER: The table will be sorted by overall descending frequency of SOC and then, within a SOC, by overall descending frequency of Preferred Term}

<sup>&</sup>lt;sup>b</sup> Counts reflect number of medical history terms that map to MedDRA.



# Table 14.1.4.1: Summary of Concomitant Medications by ATC Level 2 and Preferred Name (Safety Population) (Page 1 of xx)

| ATC Level 2 Term <sup>a</sup> Preferred Name | E-BPO 5% Cream<br>(N=xxx) |
|---|---|
| Number (%) of Subjects Reporting at Least One Concomitant Medication | xx ( xx.x%) |
| ATC Level 2 Term Preferred Name | xx ( xx.x%)<br>xx ( xx.x%) |

Note: WHO Drug Global Dictionary, Format B3, Version March 1, 2018
Concomitant medications are those used on/after the date of first application of E-BPO 5% Cream (from SGT-54-01/SGT-54-02 or SGT-54-07).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Counts reflect number of subjects reporting one or more medications that map to the WHO term. At each level of summarization (ATC Level 2 Term or Preferred Name) subjects are counted once. Percentages are based on the number of subjects in the safety population.



Table 14.2.1.1: Summary of Investigator Global Assessment at Baseline and Week 40 (Safety Population)

| | SGT-54-01/SGT-54-02 | SGT-54-01/SG-54-02 | SGT-54-07 |
|---|---|---|---|
| | Vehicle Cream | E-BPO 5% Cream | E-BPO 5% Cream |
| Investigator Global Assessment | (N=xxx) | N=xxx | (N=xxx) |
| Baseline <sup>a</sup> | | | |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 40/ET <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based on nominal visit Week 40/ET from SGT-54-07.


Table 14.2.1.2: Summary of Investigator Global Assessment at Each Evaluation (Safety Population)


| | SGT-54-01/SGT-54-02 | SGT-54-01/SG-54-02 | SGT-54-07 |
|---|---|---|---|
| | Vehicle Cream | E-BPO 5% Cream | E-BPO 5% Cream |
| nvestigator Global Assessment | (N=xxx) | (N=xxx) | N=xxx |
| Baseline <sup>a</sup> | · | | |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Veek 4 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.1.2: Summary of Investigator Global Assessment at Each Evaluation (Safety Population)


| | SGT-54-01/SGT-54-02<br>Vehicle Cream | SGT-54-01/SG-54-02<br>E-BPO 5% Cream | SGT-54-07<br>E-BPO 5% Cream |
|---|---|---|---|
| nvestigator Global Assessment | N=xxx | (N=xxx) | N=xxx |
| Week 8 <sup>b</sup> | · | | |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.1.2: Summary of Investigator Global Assessment at Each Evaluation (Safety Population)


| | G G T 5 4 0 1 / G G T 5 4 0 2 | GGT 54 01/GG 54 00 | CCT 54.05 |
|---|---|---|---|
| | SGT-54-01/SGT-54-02 | SGT-54-01/SG-54-02 | SGT-54-07 |
| | Vehicle Cream | E-BPO 5% Cream | E-BPO 5% Cream |
| Investigator Global Assessment | (N=xxx) | N=xxx | (N=xxx) |
| Week 16 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 20 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.1.2: Summary of Investigator Global Assessment at Each Evaluation (Safety Population)


| | SGT-54-01/SGT-54-02<br>Vehicle Cream | SGT-54-01/SG-54-02<br>E-BPO 5% Cream | SGT-54-07<br>E-BPO 5% Cream |
|---|---|---|---|
| nvestigator Global Assessment<br>Veek 24 <sup>b</sup> | (N=xxx) | (N=xxx) | (N=xxx) |
| n | xx | XX | XX |
| 0 - Clear | | | |
| 1 - Almost Clear | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) |
| | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) |
| 3 - Moderate | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Veek 28 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

TOOL.AN.10-01.01 Statistical Analysis Plan Template


<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.1.2: Summary of Investigator Global Assessment at Each Evaluation (Safety Population)


| | SGT-54-01/SGT-54-02<br>Vehicle Cream | SGT-54-01/SG-54-02<br>E-BPO 5% Cream | SGT-54-07<br>E-BPO 5% Cream |
|---|---|---|---|
| nvestigator Global Assessment | (N=xxx) | (N=xxx) | (N=xxx) |
| Week 32 <sup>b</sup> | (IV AAA) | (IV AAA) | (IV AAA) |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 1 - Almost Clear | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Week 36 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.1.2: Summary of Investigator Global Assessment at Each Evaluation (Safety Population)


| | GGT 54 01/GGT 54 00 | GGT 54 01/GG 54 02 | G G T . 5.4.05 |
|---|---|---|---|
| | SGT-54-01/SGT-54-02 | SGT-54-01/SG-54-02 | SGT-54-07 |
| | Vehicle Cream | E-BPO 5% Cream | E-BPO 5% Cream |
| Investigator Global Assessment | N=xxx | (N=xxx) | (N=xxx) |
| Week 40 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 44 <sup>b</sup> | | | |
| n | XX | NA | XX |
| 0 - Clear | xx ( xx.x%) | | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | | xx ( xx.x%) |
| 2 - Mild | xx (xx.x%) | | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx (xx.x%) | | xx ( xx.x%) |
| Failure | xx ( xx.x%) | | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.1.2: Summary of Investigator Global Assessment at Each Evaluation (Safety Population)


| | SGT-54-01/SGT-54-02 | SGT-54-01/SG-54-02 | SGT-54-07 |
|---|---|---|---|
| | Vehicle Cream | E-BPO 5% Cream | E-BPO 5% Cream |
| nvestigator Global Assessment | N=xxx | N=xxx | (N=xxx) |
| Week 48 <sup>b</sup> | | | |
| n | XX | NA | XX |
| 0 - Clear | xx ( xx.x%) | | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx ( xx.x%) | | xx ( xx.x%) |
| Failure | xx ( xx.x%) | | xx ( xx.x%) |
| Week 52 <sup>b</sup> | | | |
| n | XX | NA | XX |
| 0 - Clear | xx ( xx.x%) | | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | | xx ( xx.x%) |
| Achieving Clear or Almost Clear | | | |
| Success | xx (xx.x%) | | xx ( xx.x%) |
| Failure | xx ( xx.x%) | | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.2.1: Summary of RosaQoL Questionnaire Responses at Baseline and Week 40 (Safety Population)


| <b>Total Score</b> Baseline <sup>a</sup> | SGT-54-01/SGT-54-02<br>Vehicle Cream<br>(N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 40/ET <sup>b</sup> | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Absolute Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Total Score calculated from the unweighted mean of all RosaQoL questions.

Symptom Subscale Score calculated from items 2, 6, 9, 16, 17, 18, and 19.

Functional Subscale Score calculated from items 13, 15, and 21.

Emotional Subscale Score calculated from items 1, 3, 4, 5, 7, 8, 10, 11, 12, 14, and 20.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>b</sup> Table summaries based on nominal visit Week 40/ET from SGT-54-07.



Table 14.2.2.1: Summary of RosaQoL Questionnaire Responses at Baseline and Week 40 (Safety Population)


| Symptom Subscala Saara | SGT-54-01/SGT-54-02<br>Vehicle Cream<br>(N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| Symptom Subscale Score Baseline <sup>a</sup> | <u>(N-XXX)</u> | (N-XXX) | (IN=XXX) |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 40/ET <sup>b</sup> | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Absolute Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Total Score calculated from the unweighted mean of all RosaQoL questions.

Symptom Subscale Score calculated from items 2, 6, 9, 16, 17, 18, and 19.

Functional Subscale Score calculated from items 13, 15, and 21.

Emotional Subscale Score calculated from items 1, 3, 4, 5, 7, 8, 10, 11, 12, 14, and 20.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>b</sup> Table summaries based on nominal visit Week 40/ET from SGT-54-07.



Table 14.2.2.1: Summary of RosaQoL Questionnaire Responses at Baseline and Week 40 (Safety Population)


| | SGT-54-01/SGT-54-02 | SGT-54-01/SG-54-02 | SGT-54-07 |
|---|---|---|---|
| | Vehicle Cream | E-BPO 5% Cream | E-BPO 5% Cream |
| Functional Subscale Score | (N=xxx) | (N=xxx) | N=xxx |
| Baseline <sup>a</sup> | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 40/ET <sup>b</sup> | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Absolute Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Total Score calculated from the unweighted mean of all RosaQoL questions.

Symptom Subscale Score calculated from items 2, 6, 9, 16, 17, 18, and 19.

Functional Subscale Score calculated from items 13, 15, and 21.

Emotional Subscale Score calculated from items 1, 3, 4, 5, 7, 8, 10, 11, 12, 14, and 20.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>b</sup> Table summaries based on nominal visit Week 40/ET from SGT-54-07.



Table 14.2.2.1: Summary of RosaQoL Questionnaire Responses at Baseline and Week 40 (Safety Population)


| | SGT-54-01/SGT-54-02<br>Vehicle Cream | SGT-54-01/SG-54-02<br>E-BPO 5% Cream | SGT-54-07<br>E-BPO 5% Cream |
|---|---|---|---|
| Emotional Subscale Score | (N=xxx) | (N=xxx) | (N=xxx) |
| Baseline <sup>a</sup> | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 40/ET <sup>b</sup> | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Absolute Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Total Score calculated from the unweighted mean of all RosaQoL questions.

Symptom Subscale Score calculated from items 2, 6, 9, 16, 17, 18, and 19.

Functional Subscale Score calculated from items 13, 15, and 21.

Emotional Subscale Score calculated from items 1, 3, 4, 5, 7, 8, 10, 11, 12, 14, and 20.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>b</sup> Table summaries based on nominal visit Week 40/ET from SGT-54-07.



Table 14.2.2.2: Summary of RosaQoL Questionnaire Responses at Each Evaluation (Safety Population)


| Γotal Score | SGT-54-01/SGT-54-02<br>Vehicle Cream<br>(N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| Baseline <sup>a</sup> | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 12 <sup>b</sup> | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Absolute Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Total Score calculated from the unweighted mean of all RosaQoL questions.

Symptom Subscale Score calculated from items 2, 6, 9, 16, 17, 18, and 19.

Functional Subscale Score calculated from items 13, 15, and 21.

Emotional Subscale Score calculated from items 1, 3, 4, 5, 7, 8, 10, 11, 12, 14, and 20.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.2.2: Summary of RosaQoL Questionnaire Responses at Each Evaluation (Safety Population)


| otal Score<br>Yeek 24 <sup>b</sup> | SGT-54-01/SGT-54-02 Vehicle Cream (N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Absolute Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Total Score calculated from the unweighted mean of all RosaQoL questions.

Symptom Subscale Score calculated from items 2, 6, 9, 16, 17, 18, and 19.

Functional Subscale Score calculated from items 13, 15, and 21.

Emotional Subscale Score calculated from items 1, 3, 4, 5, 7, 8, 10, 11, 12, 14, and 20.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.2.2: Summary of RosaQoL Questionnaire Responses at Each Evaluation (Safety Population)


| otal Score<br>Veek 36 <sup>b</sup> | SGT-54-01/SGT-54-02 Vehicle Cream (N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Absolute Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Total Score calculated from the unweighted mean of all RosaQoL questions.

Symptom Subscale Score calculated from items 2, 6, 9, 16, 17, 18, and 19.

Functional Subscale Score calculated from items 13, 15, and 21.

Emotional Subscale Score calculated from items 1, 3, 4, 5, 7, 8, 10, 11, 12, 14, and 20.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.2.2: Summary of RosaQoL Questionnaire Responses at Each Evaluation (Safety Population)


| otal Score<br>Veek 40 <sup>b</sup> | SGT-54-01/SGT-54-02<br>Vehicle Cream<br>(N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| n | NA | XX | XX |
| Mean | | XX.X | XX.X |
| SD | | XX.XX | XX.XX |
| Median | | XX.X | XX.X |
| Min. to Max. | | xx to xx | xx to xx |
| Absolute Change from Baseline | | | |
| n | NA | XX | XX |
| Mean | | XX.X | XX.X |
| SD | | XX.XX | XX.XX |
| Median | | XX.X | XX.X |
| Min. to Max. | | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Total Score calculated from the unweighted mean of all RosaQoL questions.

Symptom Subscale Score calculated from items 2, 6, 9, 16, 17, 18, and 19.

Functional Subscale Score calculated from items 13, 15, and 21.

Emotional Subscale Score calculated from items 1, 3, 4, 5, 7, 8, 10, 11, 12, 14, and 20.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.2.2: Summary of RosaQoL Questionnaire Responses at Each Evaluation (Safety Population)


| otal Score<br>Veek 48 <sup>b</sup> | SGT-54-01/SGT-54-02 Vehicle Cream (N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| n | XX | NA | XX |
| Mean | XX.X | | XX.X |
| SD | XX.XX | | xx.xx |
| Median | XX.X | | XX.X |
| Min. to Max. | xx to xx | | xx to xx |
| Absolute Change from Baseline | | | |
| n | XX | NA | XX |
| Mean | XX.X | | XX.X |
| SD | XX.XX | | XX.XX |
| Median | XX.X | | XX.X |
| Min. to Max. | xx to xx | | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Total Score calculated from the unweighted mean of all RosaQoL questions.

Symptom Subscale Score calculated from items 2, 6, 9, 16, 17, 18, and 19.

Functional Subscale Score calculated from items 13, 15, and 21.

Emotional Subscale Score calculated from items 1, 3, 4, 5, 7, 8, 10, 11, 12, 14, and 20.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.2.2: Summary of RosaQoL Questionnaire Responses at Each Evaluation (Safety Population)


| otal Score<br>eek 52 <sup>b</sup> | SGT-54-01/SGT-54-02 Vehicle Cream (N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| n | XX | NA | XX |
| Mean | XX.X | | xx.x |
| SD | XX.XX | | xx.xx |
| Median | XX.X | | XX.X |
| Min. to Max. | xx to xx | | xx to xx |
| Absolute Change from Baseline | | | |
| n | XX | NA | XX |
| Mean | XX.X | | XX.X |
| SD | XX.XX | | XX.XX |
| Median | XX.X | | XX.X |
| Min. to Max. | xx to xx | | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Total Score calculated from the unweighted mean of all RosaQoL questions.

Symptom Subscale Score calculated from items 2, 6, 9, 16, 17, 18, and 19.

Functional Subscale Score calculated from items 13, 15, and 21.

Emotional Subscale Score calculated from items 1, 3, 4, 5, 7, 8, 10, 11, 12, 14, and 20.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat these pages for [Symptom Subscale Score, Functional Subscale Score and Emotional Subscale Score].

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.3: Summary of Erythema Assessment at Each Evaluation (Safety Population)


| | SGT-54-01/SGT-54-02 | SGT-54-01/SG-54-02 | SGT-54-07 |
|---|---|---|---|
| | Vehicle Cream | E-BPO 5% Cream | E-BPO 5% Cream |
| Rosacea Erythema Assessment | (N=xxx) | (N=xxx) | (N=xxx) |
| Baseline <sup>a</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 8 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.3: Summary of Erythema Assessment at Each Evaluation (Safety Population)


| | SGT-54-01/SGT-54-02 | SGT-54-01/SG-54-02 | SGT-54-07 |
|---|---|---|---|
| | Vehicle Cream | E-BPO 5% Cream | E-BPO 5% Cream |
| Rosacea Erythema Assessment | (N=xxx) | (N=xxx) | (N=xxx) |
| Week 12 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 16 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 20 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx = (xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.3: Summary of Erythema Assessment at Each Evaluation (Safety Population)


| Rosacea Erythema Assessment | SGT-54-01/SGT-54-02<br>Vehicle Cream<br>(N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| Week 24 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 28 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 32 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.3: Summary of Erythema Assessment at Each Evaluation (Safety Population)


| Rosacea Erythema Assessment | SGT-54-01/SGT-54-02<br>Vehicle Cream<br>(N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| Week 36 <sup>b</sup> | (IV MM) | (IV MM) | (IV MAIL) |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 40 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 44 <sup>b</sup> | | | |
| n | XX | NA | XX |
| 0 - None | xx (xx.x%) | | xx ( xx.x%) |
| 1 - Mild | xx (xx.x%) | | xx ( xx.x%) |
| 2 - Moderate | xx (xx.x%) | | xx ( xx.x%) |
| 3 - Severe | xx (xx.x%) | | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.3: Summary of Erythema Assessment at Each Evaluation (Safety Population) 

| Rosacea Erythema Assessment<br>Week 48 <sup>b</sup> | SGT-54-01/SGT-54-02 Vehicle Cream (N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| n | XX | NA | XX |
| 0 - None | xx ( xx.x%) | | xx ( xx.x%) |
| 1 - Mild | xx (xx.x%) | | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | | xx ( xx.x%) |
| Week 52 <sup>b</sup> | | | |
| n | XX | NA | XX |
| 0 - None | xx ( xx.x%) | | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.4: Summary of Telangiectasia Assessment at Each Evaluation (Safety Population)


| | SGT-54-01/SGT-54-02<br>Vehicle Cream | SGT-54-01/SG-54-02<br>E-BPO 5% Cream | SGT-54-07<br>E-BPO 5% Cream |
|---|---|---|---|
| Felangiectasia Assessment | (N=xxx) | (N=xxx) | (N=xxx) |
| Baseline <sup>a</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 8 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.4: Summary of Telangiectasia Assessment at Each Evaluation (Safety Population)


| | SGT-54-01/SGT-54-02<br>Vehicle Cream | SGT-54-01/SG-54-02<br>E-BPO 5% Cream | SGT-54-07<br>E-BPO 5% Cream |
|---|---|---|---|
| Felangiectasia Assessment | (N=xxx) | (N=xxx) | (N=xxx) |
| Week 12 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 16 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 20 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.4: Summary of Telangiectasia Assessment at Each Evaluation (Safety Population)


| | SGT-54-01/SGT-54-02<br>Vehicle Cream | SGT-54-01/SG-54-02<br>E-BPO 5% Cream | SGT-54-07<br>E-BPO 5% Cream |
|---|---|---|---|
| Felangiectasia Assessment | (N=xxx) | N=xxx | N=xxx |
| Week 24 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 28 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 32 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.4: Summary of Telangiectasia Assessment at Each Evaluation (Safety Population)


| | SGT-54-01/SGT-54-02<br>Vehicle Cream | SGT-54-01/SG-54-02<br>E-BPO 5% Cream | SGT-54-07<br>E-BPO 5% Cream |
|---|---|---|---|
| <b>Felangiectasia Assessment</b> Week 36 <sup>b</sup> | (N=xxx) | (N=xxx) | (N=xxx) |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 40 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 44 <sup>b</sup> | | | |
| n | XX | NA | XX |
| 0 - None | xx ( xx.x%) | | xx (xx.x%) |
| 1 - Mild | xx ( xx.x%) | | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | | xx ( xx.x%) |
| 3 - Severe | xx ( xx.x%) | | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.4: Summary of Telangiectasia Assessment at Each Evaluation (Safety Population)


| Гelangiectasia Assessment | SGT-54-01/SGT-54-02<br>Vehicle Cream<br>(N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| i eiangiectasia Assessment | (IN-XXX) | (IN-XXX) | (N-XXX) |
| Week 48 <sup>b</sup> | | | |
| n | XX | NA | XX |
| 0 - None | xx (xx.x%) | | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | | xx (xx.x%) |
| 3 - Severe | xx ( xx.x%) | | xx ( xx.x%) |
| Week 52 <sup>b</sup> | | | |
| n | XX | NA | XX |
| 0 - None | xx (xx.x%) | | xx ( xx.x%) |
| 1 - Mild | xx (xx.x%) | | xx ( xx.x%) |
| 2 - Moderate | xx ( xx.x%) | | xx ( xx.x%) |
| 3 - Severe | xx (xx.x%) | | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.2.5: Summary of Reoccurrence (Safety Population)

| | E-BPO 5% Cream (N=xxx) |
|---|---|
| Number of Retreatments | |
| n n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| Number of Treatment Free Days Until First Retreatment | |
| n | XX |
| Median <sup>c</sup> (days) | XX.X |
| 95% Confidence Interval <sup>c</sup> | (xx.x, xx.x) |

<sup>&</sup>lt;sup>a</sup> Number of retreatments is defined as the number of times a subject's IGA goes from clear or almost clear to mild, moderate or severe after the subject was clear or almost clear while receiving E-BPO 5% Cream.

b Number of treatment free days until first retreatment is defined as the number of days between an initial IGA assessment of clear or almost clear while the subject was receiving E-BPO 5% Cream until an IGA of mild, moderate or severe.

<sup>&</sup>lt;sup>c</sup> Median and 95% confidence intervals based on Kaplan-Meier method.



Table 14.3.0.1: Summary of Extent of Exposure (Safety Population) 

| | SGT-54-01/SGT-54-02 | SGT-54-01/SG-54-02 | SGT-54-07 |
|---|---|---|---|
| | Vehicle Cream | E-BPO 5% Cream | E-BPO 5% Cream |
| | (N=xxx) | (N=xxx) | (N=xxx) |
| otal Number of Days of Exposure | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| otal Number of Applications | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Otal Number of Non-Instructed Missed Applications <sup>a</sup> | | | |
| n | XX | XX | xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

a Non-Instructed missed applications are missed doses on the CRF with reason of "Other, specify reason". b Instructed missed applications are missed doses on the CRF with reason of "Per PI Instruction".



Table 14.3.0.1: Summary of Extent of Exposure (Safety Population) 

| Total Number of Instructed Missed Applications <sup>b</sup> | SGT-54-01/SGT-54-02<br>Vehicle Cream<br>(N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

a Non-Instructed missed applications are missed doses on the CRF with reason of "Other, specify reason". Instructed missed applications are missed doses on the CRF with reason of "Per PI Instruction".



Table 14.3.1.1: Summary of Cutaneous Safety and Tolerability Evaluations (Safety Population)


| | SGT-54-01/SGT-54-02<br>Vehicle Cream | SGT-54-01/SG-54-02<br>E-BPO 5% Cream | SGT-54-07<br>E-BPO 5% Cream |
|---|---|---|---|
| Dryness | $\underline{\hspace{1cm}(N=xxx)}$ | (N=xxx) | (N=xxx) |
| Baseline <sup>a</sup> | | | |
| n | XX | XX | XX |
| 0 – None | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| 1 – Mild | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) |
| 2 – Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx = (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 2 – Moderate | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}.\mathbf{x}\%)$ | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | XX (XX.X%) |
| Week 8 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | XX (XX.X%) | xx = (xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx = (xx.x%) | xx ( xx.x%) |
| 2 – Moderate | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}.\mathbf{x}\%)$ | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}.\mathbf{x}\%)$ | xx ( xx.x%) |
| 3 – Severe | $\mathbf{x}\mathbf{x} = (\mathbf{x}\mathbf{x}\mathbf{x}\mathbf{x}'')$ | $\mathbf{x}\mathbf{x} = (\mathbf{x}$ | $\mathbf{x}\mathbf{x} = (\mathbf{x}$ |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.3.1.1: Summary of Cutaneous Safety and Tolerability Evaluations (Safety Population)


| | SGT-54-01/SGT-54-02 | SGT-54-01/SG-54-02 | SGT-54-07 |
|---|---|---|---|
| | Vehicle Cream | E-BPO 5% Cream | E-BPO 5% Cream |
| Dryness | (N=xxx) | N=xxx | N=xxx |
| Week 12 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0-None | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 16 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0-None | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 20 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx = (xx.x%) | xx = (xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.3.1.1: Summary of Cutaneous Safety and Tolerability Evaluations (Safety Population)


| | SGT-54-01/SGT-54-02 | SGT-54-01/SG-54-02 | SGT-54-07 |
|---|---|---|---|
| | Vehicle Cream | E-BPO 5% Cream | E-BPO 5% Cream |
| Dryness | N=xxx | (N=xxx) | N=xxx |
| Week 24 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0-None | xx ( xx.x%) | xx = (xx.x%) | xx (xx.x%) |
| 1 – Mild | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx = (xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 28 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0-None | xx ( xx.x%) | xx = (xx.x%) | xx (xx.x%) |
| 1 – Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx = (xx.x%) | xx (xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 32 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx = (xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx = (xx.x%) | xx ( xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.3.1.1: Summary of Cutaneous Safety and Tolerability Evaluations (Safety Population)


| | SGT-54-01/SGT-54-02 | SGT-54-01/SG-54-02 | SGT-54-07 |
|---|---|---|---|
| | Vehicle Cream | E-BPO 5% Cream | E-BPO 5% Cream |
| Dryness | (N=xxx) | N=xxx | (N=xxx) |
| Week 36 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0-None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Week 40 <sup>b</sup> | | | |
| n | XX | XX | XX |
| 0-None | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 - Mild | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 44 <sup>b</sup> | | | |
| n | XX | NA | XX |
| 0 - None | xx ( xx.x%) | | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | | xx ( xx.x%) |
| 3 – Severe | xx = (xx.x%) | | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.3.1.1: Summary of Cutaneous Safety and Tolerability Evaluations (Safety Population)


| <b>Pryness</b><br>Veek 48 <sup>b</sup> | SGT-54-01/SGT-54-02<br>Vehicle Cream<br>(N=xxx) | SGT-54-01/SG-54-02<br>E-BPO 5% Cream<br>(N=xxx) | SGT-54-07<br>E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|---|
| n | XX | NA | XX |
| 0 - None | xx = (xx.x%) | | xx (xx.x%) |
| 1 – Mild | xx = (xx.x%) | | xx ( xx.x%) |
| 2 – Moderate | xx = (xx.x%) | | xx = (xx.x%) |
| 3 – Severe | xx ( xx.x%) | | xx (xx.x%) |
| Veek 52 <sup>b</sup> | | | |
| n | XX | NA | XX |
| 0 - None | xx ( xx.x%) | | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | | xx ( xx.x%) |
| 3 – Severe | xx = (xx.x%) | | xx = (xx.x%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Repeat these pages for [Scaling, Itching and Burning/Stinging]

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



Table 14.3.1.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population)


| | E-BPO 5% Cream (N=xxx) |
|---|---|
| Subjects Reporting Any Treatment-Emergent Adverse Event Number of Treatment-Emergent Adverse Events | xx ( xx.x%)<br>xx |
| Subjects Reporting Any Serious Treatment-Emergent Adverse Event<br>Number of Serious Treatment-Emergent Adverse Events | xx (xx.x%)<br>xx |
| Subjects Reporting Treatment-Emergent Adverse Event with Outcome of Fatal Number of Treatment-Emergent Adverse Events with Outcome of Fatal | xx ( xx.x%)<br>xx |
| Subjects Who Discontinued Study Drug Due to a Treatment-Emergent Adverse Event Number of Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug | xx (xx.x%)<br>xx |
| Subjects Who Discontinued from the Study Due to a Treatment-Emergent Adverse Event Number of Treatment-Emergent Adverse Events Leading to Discontinuation of Study | xx ( xx.x%)<br>xx |

Note: Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream. Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".


Table 14.3.1.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population)


| | E-BPO 5% Cream (N=xxx) |
|---|---|
| By Maximum Severity Severe Moderate Mild | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| By Strongest Relationship to Study Drug<br>Related<br>Not Related | xx ( xx.x%)<br>xx ( xx.x%) |
| Maximum Severity within Relationship to Study Drug Related Severe Moderate | xx ( xx.x%)<br>xx ( xx.x%) |
| Mild Not Related Severe | $\begin{array}{ccc} xx & (& xx.x\%) \\ xx & (& xx.x\%) \end{array}$ $xx & (& xx.x\%)$ |
| Moderate<br>Mild | xx ( xx.x%)<br>xx ( xx.x%) |

Note: Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream. Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".



## Table 14.3.1.2.2: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population) (Page 1 of x)

| System Organ Class <sup>a</sup> Preferred Term | E-BPO 5% Cream (N=xxx) |
|------------------------------------------------|----------------------------|
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Note: MedDRA Version 21.0

Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.



Table 14.3.1.2.3: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population)

| System Organ Class <sup>a</sup> Preferred Term | <u>Severity</u> | E-BPO 5% Cream (N=xxx) |
|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Severe<br>Moderate<br>Mild | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Severe<br>Moderate<br>Mild | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

Note: MedDRA Version 21.0.

Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.



### Table 14.3.1.2.4: Summary of Treatment-Emergent Adverse Events by Relationship to Study Drug (Safety Population) (Page 1 of xx)

| System Organ Class <sup>a</sup> Preferred Term | Relationship | E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Related<br>Not Related | xx ( xx.x%)<br>xx ( xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxxxx | Related<br>Not Related | xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

Note: MedDRA Version 21.0.

Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream. Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".



Table 14.3.1.3.1: Summary of Treatment-Emergent Adverse Event Characteristics - By Period (Safety Population)


| Subjects Reporting Any Treatment-Emergent Adverse Event<br>Number of Treatment-Emergent Adverse Events | 0-12 Weeks<br>(N=xxx)<br>xx (xx.x%)<br>xx | >12-28 Weeks<br>(N=xxx)<br>xx (xx.x%)<br>xx | >28-52 Weeks<br>(N=xxx)<br>xx (xx.x%)<br>xx | >52 Weeks<br>(N=xxx)<br>xx (xx.x%)<br>xx |
|---|---|---|---|---|
| Subjects Reporting Any Serious Treatment-Emergent Adverse Event<br>Number of Serious Treatment-Emergent Adverse Events | xx (xx.x%)<br>xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%)<br>xx |
| Subjects Reporting Treatment-Emergent Adverse Event with Outcome of Fatal Number of Treatment-Emergent Adverse Events with Outcome of Fatal | xx (xx.x%)<br>xx | xx (xx.x%) | xx (xx.x%)<br>xx | xx (xx.x%)<br>xx |
| Subjects Who Discontinued Study Drug Due to a Treatment-Emergent Adverse Event Number of Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug | xx (xx.x%)<br>xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%)<br>xx |
| Subjects Who Discontinued from the Study Due to a Treatment-Emergent Adverse Event Number of Treatment-Emergent Adverse Events Leading to Discontinuation of Study | xx (xx.x%)<br>xx | xx (xx.x%)<br>xx | xx (xx.x%)<br>xx | xx (xx.x%)<br>xx |

Note: Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.

Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".

Periods defined from date of first dose of E-BPO 5% Cream. Period >52 Weeks includes all adverse events reported after week 52 through the end of study participation.

By subject denominator for each period includes the number of subjects in the safety population completing the period or experiencing an adverse event during the period.



Table 14.3.1.3.1: Summary of Treatment-Emergent Adverse Event Characteristics – By Period (Safety Population)


| By Maximum Severity | 0-12 Weeks<br>(N=xxx) | >12-28 Weeks<br>(N=xxx) | >28-52 Weeks<br>(N=xxx) | >52 Weeks<br>(N=xxx) |
|---|---|---|---|---|
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) | xx = (xx.x%) | xx ( xx.x%) |
| Mild | xx (xx.x%) | xx ( xx.x%) | xx = (xx.x%) | xx ( xx.x%) |
| Mild | AA ( AA.A70) | AA (AA.A70) | AA (AA.A70) | AA (AA.A70) |
| By Strongest Relationship to Study Drug | | | | |
| Related | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Related | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | , | , | , | , |
| Maximum Severity within Relationship to Study Drug | | | | |
| Related | | | | |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Related | | | | |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.

Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".

Periods defined from date of first dose of E-BPO 5% Cream. Period >52 Weeks includes all adverse events reported after week 52 through the end of study participation.

By subject denominator for each period includes the number of subjects in the safety population completing the period or experiencing an adverse event during the period.



Table 14.3.1.3.2: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term – By Period (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | 0-12 Weeks | >12-28 Weeks | >28-52 Weeks | >52 Weeks |
|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | , |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once. By subject denominator for each period includes the number of subjects in the safety population completing the period or experiencing an adverse event during the period.

Note: MedDRA Version 21.0

Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.

Periods defined from date of first dose of E-BPO 5% Cream. Period >52 Weeks includes all adverse events reported after week 52 through the end of study participation.



Table 14.3.1.3.3: Summary of Treatment-Emergent Adverse Events by Severity – By Period (Safety Population)

| System Organ Class <sup>a</sup> Preferred Term | Severity | 0-12 Weeks<br>(N=xxx) | >12-28 Weeks<br>(N=xxx) | >28-52 Weeks<br>(N=xxx) | >52 Weeks<br>(N=xxx) |
|---|---|---|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxxx | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported reported severity. By subject denominator for each period includes the number of subjects in the safety population completing the period or experiencing an adverse event during the period.

Note: MedDRA Version 21.0

Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.

Periods defined from date of first dose of E-BPO 5% Cream. Period >52 Weeks includes all adverse events reported after week 52 through the end of study participation.



Table 14.3.1.3.4: Summary of Treatment-Emergent Adverse Events by Relationship to Study Drug – By Period (Safety Population)

| System Organ Class <sup>a</sup> Preferred Term | Relationship | 0-12 Weeks<br>(N=xxx) | >12-28 Weeks<br>(N=xxx) | >28-52 Weeks<br>(N=xxx) | >52 Weeks<br>(N=xxx) |
|---|---|---|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxxxx | Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Not Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxxx | Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Not Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship. By subject denominator for each period includes the number of subjects in the safety population completing the period or experiencing an adverse event during the period.

Note: MedDRA Version 21.0.

Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.

Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".

Periods defined from date of first dose of E-BPO 5% Cream. Period >52 Weeks includes all adverse events reported after week 52 through the end of study participation.



Table 14.3.1.4.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population)


| Subjects Reporting Any Serious Treatment-Emergent Adverse Event<br>Number of Serious Treatment-Emergent Adverse Events | E-BPO 5% Cream (N=xxx) xx ( xx.x%) xx |
|---|---|
| Subjects Reporting Serious Treatment-Emergent Adverse Event with Outcome of Fatal Number of Serious Treatment-Emergent Adverse Events with Outcome of Fatal | xx ( xx.x%)<br>xx |
| Subjects Who Discontinued Study Drug Due to a Serious Treatment-Emergent Adverse Event Number of Serious Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug | xx ( xx.x%)<br>xx |
| Subjects Who Discontinued from the Study Due to a Serious Treatment-Emergent Adverse Event Number of Serious Treatment-Emergent Adverse Events Leading to Discontinuation of Study | xx ( xx.x%)<br>xx |

Note: Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream. Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".



Table 14.3.1.4.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population)


| | E-BPO 5% Cream |
|----------------------------------------------------|----------------|
| | (N=xxx) |
| By Maximum Severity | (= : =====) |
| Severe | xx ( xx.x%) |
| Moderate | xx ( xx.x%) |
| Mild | xx (xx.x%) |
| By Strongest Relationship to Study Drug | |
| Related | xx (xx.x%) |
| Not Related | xx ( xx.x%) |
| | , |
| Maximum Severity within Relationship to Study Drug | |
| Related | |
| | ( 0/) |
| Severe | xx ( xx.x%) |
| Moderate | xx ( xx.x%) |
| Mild | xx (xx.x%) |
| Not Related | |
| Severe | xx (xx.x%) |
| Moderate | xx ( xx.x%) |
| Mild | xx ( xx.x%) |
| ****** | m ( mm/v) |

Note: Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream. Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".



## Table 14.3.1.4.2: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population) (Page 1 of x)

| System Organ Class <sup>a</sup> Preferred Term | E-BPO 5% Cream (N=xxx) |
|------------------------------------------------|----------------------------|
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Note: MedDRA Version 21.0

Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.



## Table 14.3.1.4.3: Summary of Serious Treatment-Emergent Adverse Events by Severity (Safety Population) (Page 1 of x)

| System Organ Class <sup>a</sup> Preferred Term | <u>Severity</u> | E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Severe<br>Moderate<br>Mild | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Severe<br>Moderate<br>Mild | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class Preferred Term) subjects are counted once under the greatest reported severity.

Note: MedDRA Version 21.0.

Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

or



### Table 14.3.1.4.4: Summary of Treatment-Emergent Serious Adverse Events by Relationship to Study Drug (Safety Population) (Page 1 of xx)

| System Organ Class <sup>a</sup> Preferred Term | Relationship | E-BPO 5% Cream<br>(N=xxx) |
|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Related<br>Not Related | xx ( xx.x%)<br>xx ( xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxxxx | Related<br>Not Related | xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

Note: MedDRA Version 21.0.

Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream. Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".



Table 14.3.1.5.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics – By Period (Safety Population)


| Subjects Reporting Any Serious Treatment-Emergent Adverse Event<br>Number of Serious Treatment-Emergent Adverse Events | 0-12 Weeks<br>(N=xxx)<br>xx (xx.x%)<br>xx | >12-28 Weeks<br>(N=xxx)<br>xx (xx.x%)<br>xx | >28-52 Weeks<br>(N=xxx)<br>xx (xx.x%)<br>xx | >52 Weeks<br>(N=xxx)<br>xx (xx.x%)<br>xx |
|---|---|---|---|---|
| Subjects Reporting Serious Treatment-Emergent Adverse Event with Outcome of Fatal Number of Serious Treatment-Emergent Adverse Events with Outcome of Fatal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx | xx | xx | xx |
| Subjects Who Discontinued Study Drug Due to a Serious Treatment-Emergent Adverse Event Number of Serious Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx | xx | xx | xx |
| Subjects Who Discontinued from the Study Due to a Serious Treatment-Emergent Adverse Event Number of Serious Treatment-Emergent Adverse Events Leading to Discontinuation of Study | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx | xx | xx | xx |

Note: Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.

Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".

Periods defined from date of first dose of E-BPO 5% Cream. Period >52 Weeks includes all adverse events reported after week 52 through the end of study participation.

By subject denominator for each period includes the number of subjects in the safety population completing the period or experiencing an adverse event during the period.



Table 14.3.1.5.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics – By Period (Safety Population)


| By Maximum Severity | 0-12 Weeks<br>(N=xxx) | >12-28 Weeks<br>(N=xxx) | >28-52 Weeks<br>(N=xxx) | >52 Weeks<br>(N=xxx) |
|---|---|---|---|---|
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}.\mathbf{x}\%)$ | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| IVIIIu | XX (XX.X/0) | XX (XX.X/0) | XX (XX.X/0) | AA (AA.A/0) |
| By Strongest Relationship to Study Drug | | | | |
| Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Maximum Severity within Relationship to Study Drug | | | | |
| Related | | | | |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Related | , | , , | , , | , |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | ` , | ` / | ` / | ` / |

Note: Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.

Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".

Periods defined from date of first dose of E-BPO 5% Cream. Period >52 Weeks includes all adverse events reported after week 52 through the end of study participation.

By subject denominator for each period includes the number of subjects in the safety population completing the period or experiencing an adverse event during the period.



Table 14.3.1.5.2: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term – By Period (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | 0-12 Weeks | >12-28 Weeks | >28-52 Weeks | >52 Weeks |
|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once. By subject denominator for each period includes the number of subjects in the safety population completing the period or experiencing an adverse event during the period.

Note: MedDRA Version 21.0

Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.

Periods defined from date of first dose of E-BPO 5% Cream. Period >52 Weeks includes all adverse events reported after week 52 through the end of study participation.



Table 14.3.1.5.3: Summary of Treatment-Emergent Serious Adverse Events by Severity – By Period (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | <u>Severity</u> | 0-12 Weeks<br>(N=xxx) | >12-28 Weeks<br>(N=xxx) | >28-52 Weeks<br>(N=xxx) | >52 Weeks<br>(N=xxx) |
|---|---|---|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxxx | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported reported severity. By subject denominator for each period includes the number of subjects in the safety population completing the period or experiencing an adverse event during the period.

Note: MedDRA Version 21.0

Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.

Periods defined from date of first dose of E-BPO 5% Cream. Period >52 Weeks includes all adverse events reported after week 52 through the end of study participation.



Table 14.3.1.5.4: Summary of Treatment-Emergent Serious Adverse Events by Relationship to Study Drug – By Period (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | Relationship | 0-12 Weeks<br>(N=xxx) | >12-28 Weeks<br>(N=xxx) | >28-52 Weeks<br>(N=xxx) | >52 Weeks<br>(N=xxx) |
|---|---|---|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxxx | Related<br>Not Related | xx (xx.x%)<br>xx (xx.x%) | , | xx ( xx.x%)<br>xx ( xx.x%) | xx (xx.x%)<br>xx (xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxxxx | Related<br>Not Related | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship. By subject denominator for each period includes the number of subjects in the safety population completing the period or experiencing an adverse event during the period.

Note: MedDRA Version 21.0.

Treatment-emergent adverse events are those events with an onset after the first application of E-BPO 5% Cream.

Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".

Periods defined from date of first dose of E-BPO 5% Cream. Period >52 Weeks includes all adverse events reported after week 52 through the end of study participation.



## Table 14.3.1.4.1: Summary of Vital Signs (Safety Population) 

| Temperature (°C) | E-BPO 5% Cream (N=xxx) |
|-----------------------|------------------------|
| Baseline <sup>a</sup> | |
| n | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| Week 12 <sup>b</sup> | |
| n | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| Change from Baseline | |
| n | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Note: Negative change values represent decrease from Baseline.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



# Table 14.3.1.4.1: Summary of Vital Signs (Safety Population) 

| Tommorotume (9C) | E-BPO 5% Cream (N=xxx) |
|----------------------|------------------------|
| Temperature (°C) | (N-XXX) |
| Week 24 <sup>b</sup> | |
| n | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| Change from Baseline | |
| n | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Note: Negative change values represent decrease from Baseline.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



# Table 14.3.1.4.1: Summary of Vital Signs (Safety Population) 

| T. (20) | E-BPO 5% Cream |
|----------------------|----------------|
| Temperature (°C) | (N=xxx) |
| Week 36 <sup>b</sup> | |
| n | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| Change from Baseline | |
| n | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Note: Negative change values represent decrease from Baseline.

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



## Table 14.3.1.4.1: Summary of Vital Signs (Safety Population) 

| Temperature (°C) | E-BPO 5% Cream (N=xxx) |
|----------------------|------------------------|
| Week 48 <sup>b</sup> | |
| n | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| Change from Baseline | |
| n | XXX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the baseline value from SGT-54-01/SGT-54-02.

Note: Negative change values represent decrease from Baseline.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Repeat these pages for [Respiratory Rate (breaths/min), Systolic Blood Pressure (mmHg), Diastolic Blood Pressure (mmHg) and Heart Rate (beats/min)]

<sup>&</sup>lt;sup>b</sup> Table summaries based analysis visits, representing time from first dose of E-BPO 5% Cream.



#### 13. INDEX OF PLANNED LISTINGS

| Listing 16.1.7: Enrollment | 98 |
|---|---|
| Listing 16.2.1.1: End of Study Information | 99 |
| Listing 16.2.2.1: Inclusion/Exclusion Criteria | 100 |
| Listing 16.2.2.2: Screen Failure | 101 |
| Listing 16.2.2.3: Protocol Deviations | 102 |
| Listing 16.2.3: Analysis Populations | 103 |
| Listing 16.2.4.1: Subject Demographic Information | 104 |
| Listing 16.2.4.2.1: Unique Medical/Surgical History Coded to MedDRA System Organd Preferred Terms | _ |
| Listing 16.2.4.2.2: Medical/Surgical History | 106 |
| Listing 16.2.4.3.1: Unique Medication Names Coded to WHO Drug Global Dictional Level 2 Terms and Preferred Names | • |
| Listing 16.2.4.3.2: Prior and Concomitant Medications | 108 |
| Listing 16.2.4.4.1: Unique Procedure/Therapy Names Coded to MedDRA System O and Preferred Terms | _ |
| Listing 16.2.4.4.2: Prior and Concomitant Procedures/Therapies | 110 |
| Listing 16.2.5.1: Study Visit Compliance | 111 |
| Listing 16.2.5.2: Subject Dosing Compliance | 112 |
| Listing 16.2.5.3: Subject Dosing | 113 |
| Listing 16.2.5.4: Study Medication Dispensation | 114 |
| Listing 16.2.5.5: Study Medication Accountability Log | 115 |
| Listing 16.2.6.1: Investigator Global Assessment | 116 |
| Listing 16.2.6.2: Inflammatory Lesion Counts | 117 |
| Listing 16.2.6.3.1: RosaQoL Descriptions | 118 |
| Listing 16.2.6.3.1: RosaQoL Descriptions | 119 |
| Listing 16.2.6.3.2: RosaQoL | 120 |
| Listing 16.2.6.3.3: RosaQoL Subscales Scores | 121 |
| Listing 16.2.6.4: Erythema Severity/Telangiectasia Assessments | 122 |
| Listing 16.2.7.1: Cutaneous Safety and Tolerability Assessments | 123 |



| Listing 16.2.7.2.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms | 124 |
|---|---|
| Listing 16.2.7.2.2: Pre-Treatment Adverse Events | 125 |
| Listing 16.2.7.2.3: Treatment-Emergent Adverse Events | 126 |
| Listing 16.2.7.2.4: Serious Adverse Events | 127 |
| Listing 16.2.7.2.5: Subjects Who Prematurely Discontinued Study and/or Discontinued Study Drug Due to Adverse Events | • |
| Listing 16.2.8.1: Urine Pregnancy Tests | 129 |
| Listing 16.2.8.1: Urine Pregnancy Tests. Listing 16.2.8.2: Physical Examination | |

### Listing 16.1.7: Enrollment (Page xx of yy)

| Subject | Age/Sex | Eval | Enrollment Date | Date of Last Application<br>From SGT-54-01/02 Study | Prior Treatment From SGT-54-01/02 Study |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxx | xxxxxxxxx | xxxxxxx xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxx | xxxxxxxxx | xxxxxxx xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxx | xxxxxxxx | xxxxxxx xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxx | xxxxxxxxx | xxxxxx xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxx | xxxxxxxxx | xxxxxx xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxx | xxxxxxxxx | xxxxxx xxxxx |
| xxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxx | xxxxxxxxx | xxxxxx xxxxx |
| xxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxx | xxxxxxxxx | xxxxxx xxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject.

### Listing 16.2.1.1: End of Study Information (Page xx of yy)

| | | | | | <del> </del> | | |
|---|---|---|---|---|---|---|---|
| Subject | Age/Sex | Eval | Date of<br>First<br>Application | Date of<br>Last<br>Application | Date of Study<br>Completion/<br>Discontinuation<br>(Day) <sup>1</sup> | Did Subject<br>Complete<br>the Study | Primary Reason<br>for Study Discontinuation |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxxxx | xxx | |
| xxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxxxx | xx | xxxxxx xxxxx |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxxxxx | xx | **** ** ******** ******* *** ** ******* |
| | | | | | | | xxxxx xxxxx xxxxx xxx xxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

#### Listing sorted by Subject.

If Primary Reason for Study Discontinuation is Lost to Follow-Up, Protocol Violation, Withdrawal by Subject, or Other, the reason specification will be included following a colon (for example, WITHDRAWAL BY SUBJECT: xxxxx)

<sup>1</sup> Day is calculated as date - date of first application of E-BPO 5% Cream (from SGT-54-01/SGT-54-02 or SGT-54-07) for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.

Listing 16.2.2.1: Inclusion/Exclusion Criteria (Page xx of yy)

| Subject | Age/Sex | Eval | Criterion Failed | Description |
|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxx | xxxxx xxx xx xxxxxxx xxxx xxxxxxxxxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxx | ***** *** ** ******* **** ************* |
| xxxxxx | xxxx | xxxxxxxx | xxxxx | ***** *** ** ******* **** ************* |
| | | | xxxxx | ***** *** ** ******* **** ************* |
| | | | xxxxx | xxxxx xxx xx xxxxxxxx xxxx xxxxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject and Criterion Failed.

### Listing 16.2.2.2: Screen Failure (Page xx of yy)

| Subject | Age/Sex | Eval | Date of<br>Screen Failure | Reason for Screen Failure |
|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | ***** *** ** ******* **** *********** |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | ***** *** ** ******* *** ************** |
| xxxxx | xxxx | xxxxxxxx | xxxxxxxxx | ***** *** ** ******* **** ************* |
| | | | xxxxxxxx | ***** *** ** ******* **** ************* |
| | | | xxxxxxxxx | ***** *** ** ******* **** ************ |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject.

### Listing 16.2.2.3: Protocol Deviations (Page xx of yy)

| Subject | Age/Sex | Eval | Deviation | Date (Day <sup>1</sup> ) |
|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxx x xxxxxxx xxx xx xxxxx xxxxx xxx xxx xx xx xxxx | xxxxxxxxxxxx |
| | | | xxxxxx xxx xx xxxxxx xxxxxx xxx xxx xx | xxxxxxxxxxxx |
| | | | xxxxxx x xxxxxxxx | |
| xxxxx | xxxx | xxxxxxxx | xxxxxx xxx xx xxxxxx xxxxxx xxx xxx xx | xxxxxxxxxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxx xxx xx xxxxxx xxxxx xxx xxx xx | xxxxxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject and Date.

<sup>1</sup> Day is calculated as date - Baseline visit date from SGT-54-07 for dates prior to Baseline visit. Otherwise, day is calculated as date - Baseline date + 1 for dates on or after Baseline visit.

### Listing 16.2.3: Analysis Populations (Page xx of yy)

| Subject | Age/Sex | Population | Included | Reason(s) Excluded |
|---------|---------|------------|----------|----------------------------|
| xxxxx | xxxx | Safety | xxx | |
| xxxxx | xxxx | Safety | xxx | |
| xxxxx | xxxx | Safety | xx | xxxxxxxxxx xxxxxx xxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject and Population (as ordered above).

Listing 16.2.4.1: Subject Demographic Information (Page xx of yy)

| Subject | Eval | B: Date of Birth<br>A: Age<br>S: Sex | R: Race<br>E: Ethnicity | C: Childbearing Potential<br>M: Method of Birth Control | Informed Consent Date |
|---|---|---|---|---|---|
| xxxxx | XXXXXXXX | B: xxxx-xx-xx<br>A: xx<br>S: xxxxx | R: xxxxxx xxxxxxxx | C: xxx<br>M: xxxxxxxxx xxxxxxxxx<br>xxxxxxxxxxx | xxxx-xx-xx |
| XXXXX | xxxxxxxx | B: xxxx-xx-xx<br>A: xx<br>S: xxxx | R: xxxxx<br>E: xxxxxxxx xx xxxxxx | C: xx<br>M: | xxxx-xx-xx |
| xxxxx | xxxxxxxx | B: xxxx-xx-xx<br>A: xx<br>S: xxxxx | R: xxxxx<br>E: xxxxxxxx xx xxxxxx | C: xxx<br>M: xxxxxxxx xxxxxxxxxxxx | xxxx-xx-xx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject.

Listing 16.2.4.2.1: Unique Medical/Surgical History Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Medical/Surgical History Verbatim Term |
|---|---|---|
| xxxx xxx xxxxxxxx xxxxxx xxxxxxxx | xxxxxxx | xxxxxx |
| | xxxx xxxxxxxx xxxxxxxx | xxxx xxxxxxxxx xxxxxx |
| xxxxxxxxx xxx xxxxxxxxxx | xxxxxxxxx | xxxxxxxxx |
| | xxxxxxxxxxx | xxxxxxxxxxx x xxxx xxx xxx |
| | | ************ ** ***** ** **** **** |

Note: System Organ Class and Preferred Term map to MedDRA (Version 21.0).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by System Organ Class, Preferred Term, and Verbatim Term.

### Listing 16.2.4.2.2: Medical/Surgical History (Page xx of yy)

| Subject | Age/Sex | Eval | Medical/Surgical History<br>Verbatim Term | S: MedDRA System Organ Class P: MedDRA Preferred Term | S: Onset Date<br>E: End Date |
|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxx | xxxxxxx | S: xxxx xxx xxxxxxxxxx xxxxxx xxxxxxxx<br>P: xxxxxxx | S: xxxx<br>E: |
| | | | ****** ** ******** ******* | S: xxxxxx xxxxxx xxxxxxxx<br>P: xxxxxxxx xxxxx xxxxxxx | S: xxxx<br>E: xxxxxxx |
| XXXXX | xxxx | xxxxxxx | xxxxxxx | S: xxxx xxx xxxxxxxxxxx xxxxxx xxxxxxxx<br>P: xxxxxxx | S: xxxx<br>E: |
| XXXXX | xxxx | xxxxxxx | xxxxxxx | S: xxxx xxx xxxxxxxxxxx xxxxxx xxxxxxxx<br>P: xxxxxxx | S: xxxx<br>E: |
| XXXXX | xxxx | xxxxxxx | xxxxxx | S: xxxx xxx xxxxxxxxxxx xxxxxx xxxxxxxx<br>P: xxxxxxx | S: xxxx<br>E: |
| | | | xxxxxxxxxxxxx | S: xxxxxx xxxxx xxxx<br>P: xxxx xxxxxxxxxx | S: xxxxxxxxx<br>E: xxxxxxxx |


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Rosacea Diagnosis (all Rosacea MH will appear first), Onset Date, End Date, Verbatim Term

Listing 16.2.4.3.1: Unique Medication Names Coded to WHO Drug Global Dictionary ATC Level 2 Terms and Preferred Names (Page xx of yy)

| WHO ATC Level 2 Term | WHO Preferred Name | Medication Verbatim Term | I: Indication<br>T: Route |
|---|---|---|---|
| xxxxxxxxxxx | xxxxxxxxxxx | xxxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |
| | | xxxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |
| xxxxxxxxxx | xxxxxxxxxxx | xxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |
| | | xxxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |

Note: ATC Level 2 Term and Preferred Name map to WHO Drug Global Dictionary, Format B3, Version March 1, 2018.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by ATC Level 2 Term, Preferred Name, Medication Verbatim Term, Indication, and Route.

### Listing 16.2.4.3.2: Prior and Concomitant Medications (Page xx of yy)

| S: Subject | A: ATC Level 2 Term | S: Start Date (Day) 1 | I: Indication | |
|---|---|---|---|---|
| A: Age/Sex | P: Preferred Name | E: End Date (Day) 1 | D: Dose | F: Frequency |
| E: Eval | M: Medication Name | P: Prior/Concomitant | U: Units | T: Route |
| S: xxxxxx | A: xxxxxxxx xxx xxxxxxxxx | S: xxxxxxxxxxxxxx | I: xxxxxxx | F: xxx |
| A: xxxx | P: xxxxxxxxxx xxxxxx xxxxxxx xxx xxx xxx | E: xxxxxxxxxxxxxx | D: xx | T: xxxxxxxxxxxxxx |
| E: xxxxxxxx | M: XXXXXX XXXXXXXXX | P: xxxxxxxxxxxxxxxxx | xx U: xxxxxxxxxx | |
| | A: xxxxxxx xx xxxxxxxx | S: xxxxxxxxxxxxxx | I: xxxxxxx | F: xx |
| | P: xxxxxxxxxx xxxxxx xxx | E: xxxxxxxxxxxxxx | D: xx | T: xxxxx |
| | M: xxxxxx xxxxxxxxx | P: xxxxx | U: xxxxxxxx | |
| S: xxxxxx | A: xxxxxxxxx xxx xxxxxxxxxx | S: xxxxxxxxxxxxxx | I: xxxxxxx | F: xxx |
| A: xxxx | P: xxxxxxxxx xxxxxx xxxxxx xxx xxx xxx x | E: xxxxxxxxxxxxxx | D: xx | T: xxxxxxxxxxxxx |
| E: xxxxxxxx | M: XXXXXX XXXXX XXXXXXXX | P: xxxxxxxxxxxxxxxxxx | xx U: xxxxxxxxxxx | |
| | A: xxxxxxx xx xxxxxxxx | S: xxxxxxxxxxxxxx | I: xxxxxxx | F: xx |
| | P: xxxxxxxxx xxxxxx xxx | E: xxxxxxxxxxxxxx | D: xx | T: xxxxx |
| | M: xxxxxx xxxxxxxx | P: xxxxx | U: xxxxxxxx | |

Note: ATC Level 2 Term and Preferred Name map to WHO Drug Global Dictionary, Format B3, Version March 1, 2018.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, Medication Name, Indication, Route, Frequency. If the Route is Topical, then the area treated is presented within parenthesis (T: Topical (specify area)).

Day is calculated as date - date of first application of E-BPO 5% Cream (from SGT-54-01/SGT-54-02 or SGT-54-07) for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.
Listing 16.2.4.4.1: Unique Procedure/Therapy Names Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Procedure/Therapy Verbatim Term | Indication |
|---|---|---|---|
| xxxxxxxxxxx | xxxxxxxxxxxx | xxxxxxx xx xxxxx | xxxxxxxxxx |
| | | xxxxxxxx | XXXXX XX XXXX |
| xxxxxxxxxxx | xxxxxxxxxxx | xxxxxxx | xxxxxxx |
| | | | XXXXXXXXX |
| | | xxxxxxxx | xxxxxxxxxx |
| xxxxx xxx xx xxxxxxx | xxxxxx xxxxxx xxxx | xxxxxxx xxxxxx | xxxxxxx xxxxxxx xx xx xxxxx |


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by System Organ Class, Preferred Term, Verbatim Term, and Indication.

Listing 16.2.4.4.2: Prior and Concomitant Procedures/Therapies (Page xx of yy)

| | | | S: MedDRA System Organ Class | S: Start Date (Day) 1 | |
|---|---|---|---|---|---|
| | | | P: MedDRA Preferred Term | E: End Date (Day) 1 | I: Indication |
| Subject | Age/Sex | Eval | M: Procedure/Therapy Name | P: Prior/Concomitant | A: Anatomical Area Treated |
| xxxxx | xxxx | xxxxxxx | S: xxxxxx xxx xxxxxxx xxxxxxx | S: xxxxxxxxxxxxxxxx | I: xxxxx xxxxxxx |
| | | | P: xxxxxxxxxx xxxxxxxx xxxxxxx | E: xxxxxxxxxxxxxxxx | A: |
| | | | M: xxxxxxx xxxxx xxxxxx xxxxxxx | P: xxxxxxxxxxxxxxx | |
| xxxxx | XXXX | xxxxxxx | S: xxxxxxx xxx xxxxxxx xxxxxxxx | S: xxxxxxxxxxxxxxxx | I: xxxxx xxxxxxx |
| | | | P: xxxxxxxxxx xxxxxxxx xxxxxxx | E: xxxxxxxxxxxxxxx | A: |
| | | | M: xxxxxx xxxxx xxxxxx xxxxxx | P: xxxxxxxxxxxxxxxx | |
| xxxxx | XXXX | xxxxxxx | S: xxxxxxx xxx xxxxxxxx xxxxxxxx | S: xxxxxxxxxxxxxxxx | I: xxxxx xxxxxxx |
| | | | P: xxxxxxxxxx xxxxxxxx xxxxxxx | E: xxxxxxxxxxxxxxxx | A: |
| | | | M: xxxxxxx xxxxx xxxxxx xxxxxx | P: xxxxxxxxxxxxxxxx | |
| | | | S: xxxxxx xxxxxxx xxxx | S: xxxxxxxxxxxxxxxx | I: xxxxxxxx xxxxx xx xx |
| | | | P: xxx xxxxxxxxx xxxxxxx | E: xxxxxxxxxxxxxxx | A: xxxxxxxxx |
| | | | M: xxxxxx xxxxxxx | P: xxxxxxxxxxxxxxxx | |
| | | | S: xxxxxx xxxxxxx xxxx | S: xxxxxxxxxxxxxxxx | I: xxxxxxxx xxxx xx xx |
| | | | P: xxx xxxxxxxxx xxxxxxx | E: xxxxxxxxxxxxxxx | A: xxxxxxxxx |
| | | | M: xxxxxx xxxxxxx | P: xxxxxxxxxxxxxxxx | |


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, Procedure/Therapy Name, and Indication.

<sup>1</sup> Day is calculated as date - date of first application of E-BPO 5% Cream (from SGT-54-01/SGT-54-02 or SGT-54-07) for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.

Listing 16.2.5.1: Study Visit Compliance (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | SGT-54-07<br>Analysis Visit | Visit<br>Date | $\mathtt{Day}^1$ | Within<br>Study<br>Window <sup>2</sup> | Reason Screening<br>And Baseline Visit<br>Occurred on<br>Different Days | Reason for<br>Unscheduled Visi |
|---|---|---|---|---|---|---|---|---|---|
| XXXXX | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | | | | |
| | | | xxxxxxx | xxxx x | xxxxxxxxx | | | xxxxxx xxx xx | |
| | | | xxxx x | xxxx x | xxxxxxxxx | | | | |
| | | | xxxx x | xxxx x | xxxxxxxxx | | | | |
| | | | xxxx xx | xxxx x | xxxxxxxxx | | | | |
| | | | XXXX XX | xxxx x | xxxxxxxxx | | | | |
| | | | XXXX XX | xxxx x | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | xxxx x | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | xxxx x | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | xxxx x | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | xxxx x | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XXXXX | xxxx x | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XX | XXX | | xxxxxxxxxxxx |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XX | XXX | | XXXXXXXXXXXX |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XX | XXX | | XXXXXXXXXXXX |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XX | XXX | | |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XX | XXX | | |

Day is calculated as date - Baseline date from SGT-54-07 for dates prior to Baseline visit. Otherwise, day is calculated as date - Baseline date + 1 for dates on or after Baseline visit. Day is only calculated for visits occurring in SGT-54-07.

Listing sorted by Subject and Visit Number.

<sup>&</sup>lt;sup>2</sup> Determined by protocol-specified visit window for scheduled visits after Baseline. Only assessed for visits occurring in SGT-54-07.

# Listing 16.2.5.2: Subject Dosing Compliance (Page xx of yy)

| xxxxx xxxx<br>xxxxx xxxx | Age/Sex | Eval | Date of First<br>Application | Date of Last<br>Application | Number of<br>Days of<br>Exposure | Total<br>Number of<br>Applications | Number of<br>Instructed<br>Missed<br>Applications <sup>1</sup> | Number of<br>Non-Instructed<br>Missed<br>Applications <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | XXXX | xxxxxxx | xxxxxxxx | xxxxxxxxx | xx | xxx | xx | xx |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxxx | xxxxxxxxx | xx | xxx | xx | xx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject.

The number instructed missed applications is the total number of missed doses on the CRF with reason "Per PI Instruction".

The number of non-instructed missed applications is the total number of missed doses on the CRF with reason of "Other, specify". reason".

# Listing 16.2.5.3: Subject Dosing (Page xx of yy)

| xxxxx xxx | Age/Sex | Eval | Study Interval | Start Date | End Date | Number of Doses<br>Applied¹ or Number<br>Of Doses Applied<br>Each Day of the<br>Date Span² | Reason Subject<br>Did Not Dose<br>or Dosed More<br>Than Once Per Day <sup>2</sup> |
|---|---|---|---|---|---|---|---|
| | | | 54 01 Direct to Took Door Takeway | | | | |
| XXXXXX | XXXX | XXXXXXX | 54-01 First to Last Dose Interval | XXXXXXXXX | XXXXXXXXX | | |
| | | | 54-01 Dosing Deviation | XXXXXXXXX | XXXXXXXXX | | |
| | | | 54-01 Dosing Deviation | XXXXXXXXX | XXXXXXXXX | | |
| | | | 54-01 Dosing Deviation 54-07 Dosing Interval | XXXXXXXXX | XXXXXXXXX | | |
| | | | 54-07 Dosing Interval | XXXXXXXXXX | XXXXXXXXXX | | XXX XX XXXXXXXX |
| | | | 54-07 Dosing Interval | XXXXXXXXX | XXXXXXXXXX | | xxx xx xxxxxxxx |
| | | | 54-07 Dosing Interval | XXXXXXXXXX | XXXXXXXXXX | | *** ** ******* |
| | | | 54-07 Dosing Interval | XXXXXXXXXX | XXXXXXXXXX | | xxx xx xxxxxxxx |
| | | | 54-07 Dosing Interval | XXXXXXXXXX | XXXXXXXXX | | AAA AA AAAAAAAA |
| xxxxx | xxxx | xxxxxxx | 54-01 First to Last Dose Interval | xxxxxxxxx | xxxxxxxxx | | |
| | | | 54-01 Dosing Deviation | xxxxxxxxx | xxxxxxxxx | x | |
| | | | 54-01 Dosing Deviation | xxxxxxxxx | xxxxxxxxx | х | |
| | | | 54-01 Dosing Deviation | xxxxxxxxx | xxxxxxxxx | x | |
| | | | 54-01 Dosing Deviation | xxxxxxxxx | xxxxxxxxx | X | |
| | | | 54-01 Dosing Deviation | XXXXXXXXX | xxxxxxxxx | x | |
| | | | 54-07 Dosing Interval | XXXXXXXXX | XXXXXXXXX | X | xxx xx xxxxxxxx |
| | | | 54-07 Dosing Interval | xxxxxxxxx | xxxxxxxxx | X | |
| xxxxx | xxxx | xxxxxxx | 54-07 Dosing Interval | xxxxxxxxx | xxxxxxxxx | X | xxx xx xxxxxxxx |
| | | | 54-07 Dosing Interval | XXXXXXXXX | XXXXXXXXX | X | |
| | | | 54-07 Dosing Interval | XXXXXXXXX | XXXXXXXXX | Х | xxx xx xxxxxxxx |
| | | | 54-07 Dosing Interval | XXXXXXXXX | XXXXXXXXX | Х | |
| | | | 54-07 Dosing Interval | XXXXXXXXX | XXXXXXXXX | Х | xxx xx xxxxxxxx |
| | | | 54-07 Dosing Interval | XXXXXXXXX | XXXXXXXXX | Х | |
| | | | 54-07 Dosing Interval | XXXXXXXXX | xxxxxxxxx | X | xxx xx xxxxxxxx |

<sup>&</sup>lt;sup>1</sup> From SGT-54-01 or SGT-54-02

Note: Dosing from the SGT-54-01 or 54-02 study was pulled forward for only subject who received E-BPO 5% Cream in the Phase 3 study.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

### Listing sorted by Subject and Start Date of Dosing Interval.

<sup>&</sup>lt;sup>2</sup> From SGT-54-7

Listing 16.2.5.4: Study Medication Dispensation (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of<br>Dispensation | Pump Number<br>Assigned | Instructions Given to the Subject<br>by the Investiator Regarding<br>When to Apply the Study Product | Reason Why a New<br>Pump Was Not<br>Dispensed |
|---|---|---|---|---|---|---|---|
| XXXXX | xxxx | xxxxxxx | xxxxxxx | xxxxxxxxx | xxxx | ********* | |
| | | | xxxx x | XXXXXXXXX | XXXX | XX XXXX XXXXXX XX X X XXXXXX XX | |
| | | | xxxx x | XXXXXXXXX | XXXX | XXXXXXX XXXXXXXXX XXXX XX X X XXXX XX | |
| | | | xxxx x | XXXXXXXXX | XXXX | XXXX X XXX | |
| | | | xxxx x | XXXXXXXXX | XXXX | xxxx xx xxxx xxxxxxx xx x x xxxxxxxx | |
| | | | xxxx x | XXXXXXXXX | XXXX | x xxxxx xxx xx | |
| | | | xxxx x | XXXXXXXXX | XXXX | | |
| | | | XXXX X | XXXXXXXXX | XXXX | xxxxxxxxx xxxx xx x x xxxx xxxxx | |
| XXXXX | xxxx | xxxxxxx | xxxxxxx | xxxxxxxxx | xxxx | xxxxxx | |
| | | | XXXX X | XXXXXXXXX | XXXX | XX XXXX XXXXXXX XX X X XXXXXX XXXXXX | |
| | | | XXXX X | XXXXXXXXX | XXXX | XXXXXXXXX XXXX XX X X XXXX XXXXX | |
| | | | XXXX X | XXXXXXXXX | XXXX | XXXX X XXX | |
| | | | XXXX X | XXXXXXXXX | XXXX | XXXX XX XXXX XXXXXXX XX X XXXXXX | |
| | | | XXXX X | XXXXXXXXX | XXXX | XXXXX X XXXXX XXX XX | |
| | | | XXXX X | XXXXXXXXX | XXXX | | |
| | | | XXXX X | XXXXXXXXX | XXXX | XXXXXXXXX XXXX XX X X XXXX XXXXX | |
| | | | XXXX X | XXXXXXXXX | XXXX | XXXX XX XXXX XXXXXXX XX X X XXXXXXX | |
| | | | XXXX X | XXXXXXX | | | X XXXXX XXXXX |
| | | | | | | | xxxxxxxx xx<br>xxx x xxx xxx |
| | | | xxxx x | xxxxxxxxx | XXXX | XXXX XX XXXX | |
| | | | xxxx x | XXXXXXXXX | XXXX | XXXXXXXXX XXXX XX X X XXXX XXXXX | |
| | | | xxxx x | xxxxxxxxx | XXXX | XXXX XX XXXX XXXXXXX XX X X XXXXXX XXXXX | |
| | | | xxxx x | xxxxxxxxx | XXXX | x xxxxx xxx xx | |
| | | | xxxx x | XXXXXXXXX | XXXX | XXXXXX XXXXX XX X X XXXXX XXXX XXX | |
| | | | xxxx x | XXXXXXXXX | XXXX | XXXXXXXXX XXXX XX X X XXXX XXXXX | |

Note to programmers: If a pump was not dispensed, NOT DONE will print in the date column. Listing sorted by Subject and Visit Number.

Listing 16.2.5.5: Study Medication Accountability Log (Page xx of yy)

| | | | Pump | Dispe | nsing | Ret <sup>-</sup> | urn | Amount |
|---|---|---|---|---|---|---|---|---|
| Subject | Age/Sex | Eval | Number | Date | Weight (g) | Date | Weight (g) | Used (g) |
| xxxxx | xxxx | xxxxxxx | xxxx | xxxxxxxxx | xxxx | xxxxxxxxx | xxxx | xxxx |
| | | | XXXX | xxxxxxxxx | XXXX | xxxxxxxxx | XXXX | XXXX |
| | | | XXXX | XXXXXXXXX | XXXX | XXXXXXXXX | XXXX | XXXX |
| | | | XXXX | XXXXXXXXX | XXX | XXXXXXXXX | XXXX | XXXX |
| | | | XXXX | XXXXXXXXX | XXXX | XXXXXXXXX | XXXX | XXXX |
| | | | XXXX | XXXXXXXXX | XXXX | XXX XXXX | | XXXX |
| | | | XXXX | XXXXXXXXX | XXXX | XXXXXXXXX | XXXX | XXXX |
| | | | XXXX | XXXXXXXXX | XXXX | XXXXXXXXX | XXXX | XXXX |
| XXXXX | XXXX | xxxxxxx | XXXX | xxxxxxxxx | xxxx | xxxxxxxxx | xxxx | XXXX |
| | | | XXXX | XXX XXXX | | | | |
| | | | XXXX | XXXXXXXXX | XXXX | XXXXXXXXX | XXXX | XXXX |
| | | | XXXX | xxxxxxxxx | XXXX | XXXXXXXXX | XXXX | XXXX |
| xxxxx | xxxx | xxxxxxx | xxxx | xxxxxxxxx | xxxx | xxxxxxxxx | xxxx | xxxx |
| | | | XXXX | xxxxxxxxx | XXXX | XXXXXXXXX | XXXX | XXXX |
| | | | XXXX | xxxxxxxxx | XXXX | xxxxxxxxx | XXXX | XXXX |
| | | | XXXX | xxxxxxxxx | XXXX | XXXXXXXXX | XXXX | XXXX |

Listing 16.2.6.1: Investigator Global Assessment (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | SGT-54-07<br>Analysis Visit | Date of<br>Assessment | Evaluator<br>Initials | Result |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | XXX | xxxxxxxxx |
| AAAAAA | AAAA | AAAAAAA | XXXX X | XXXX X | XXXXXXXXXX | XXX | XXXXXXXXXX |
| | | | XXXX X | XXXX X | XXXXXXXXXX | XXX | XXXXXXXXXX |
| | | | XXXX XX | XXXX X | XXXXXXXXXX | XXX | XXXXXXXXXX |
| | | | XXXX XX | XXXX X | XXXXXXXXXX | XXX | XXXXXXXXXX |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XXX | XXXXXXXXX |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XXX | XXXXXXXXX |
| | | | xxxx xx | XXXX X | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | XXXX XX | xxxx x | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | xxxx xx | XXXX X | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | XXXX XXXXX | XXXX X | xxxxxxxxx | XXX | xxxxxxxxx |
| XXXXX | XXXX | XXXXXXX | XXXXXXXX | xxxxxxxx | XXXXXXXXX | XXX | XXXXXXXXX |
| | | | XXXX X | XXXX X | XXXXXXXXX | XXX | XXXXXXXXX |
| | | | XXXX X | XXXX X | XXXXXXXXX | XXX | XXXXXXXXX |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XXX | XXXXXXXXX |
| | | | XXXX XXXXX | XXXX X | XXXXXXXXX | XXX | XXXXXXXXX |

Listing sorted by Subject and Visit Number

Listing 16.2.6.2: Inflammatory Lesion Counts (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | SGT-54-07<br>Analysis Visit | Date of<br>Assessment | Evaluator<br>Initials | Papules | Pustules | Total<br>Inflammatory<br>Lesion Count | Nodules/<br>Cysts |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | XXX | XX | XX | XX | X |
| | | | XXXX X | XXXX X | xxxxxxxxx | XXX | XX | XX | XX | Х |
| | | | XXXX X | XXXX X | xxxxxxxxx | XXX | XX | XX | XX | х |
| | | | XXXX XX | XXXX X | xxxxxxxxx | XXX | XX | XX | XX | Х |
| | | | XXXX XX | xxxx x | xxxxxxxxx | XXX | XX | XX | XX | Х |
| | | | XXXX XX | XXXX X | xxxxxxxxx | XXX | XX | XX | XX | Х |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XXX | XX | XX | XX | Х |
| | | | XXXX XX | xxxx x | XXXXXXXXX | XXX | XX | XX | XX | X |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XXX | XX | XX | XX | X |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XXX | XX | XX | XX | X |
| | | | xxxx xxxxx | XXXX X | xxxxxxxxx | xxx | XX | xx | XX | X |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | XXX | XX | XX | xx | Х |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | XXX | XX | XX | XX | Х |
| xxxxx | XXXX | xxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | xxx | xx | xx | xx | Х |
| | | | XXXX X | XXXX X | XXXXXXXXX | XXX | XX | XX | XX | X |
| | | | XXXX X | XXXX X | XXXXXXXXX | XXX | XX | XX | XX | X |
| | | | XXXX XX | XXXX X | XXXXXXXXX | XXX | XX | XX | XX | X |
| | | | XXXX XXXXX | XXXX X | XXXXXXXXX | XXX | XX | XX | XX | X |

Listing sorted by Subject and Visit Number

# Listing 16.2.6.3.1: RosaQoL Descriptions (Page xx of yy)

| Number | RosaQoL Question |
|--------|-------------------------------------------------------------------|
| 1 | I worry that my rosacea may be serious |
| 2 | My rosacea burns or stings |
| 3 | I worry about getting scars from my rosacea |
| 4 | I worry that my rosacea may get worse |
| 5 | I worry about side effects from rosacea medications |
| 6 | My rosacea is irritated |
| 7 | I am embarrassed by my rosacea |
| 8 | I am frustrated by my rosacea |
| 9 | My rosacea makes my skin sensitive |
| 10 | I am annoyed by my rosacea |
| 11 | I am bothered by the appearance of my skin (redness, blotchiness) |
| 12 | My rosacea makes me feel self-conscious |
| 13 | I try to cover up my rosacea (with make-up) |
| 14 | I am bothered by persistence/reoccurrence of my rosacea |
| 15 | I avoid certain foods or drinks because of my rosacea |
| 16 | My skin feels bumpy (uneven, not smooth, irregular) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

# Listing 16.2.6.3.1: RosaQoL Descriptions (Page xx of yy)

| Number | RosaQoL Question |
|---|---|
| 17 | My skin flushes |
| 18 | My skin gets irritated easily (cosmetics, aftershaves, cleansers) |
| 19 | My eyes bother me (feels dry or gritty) |
| 20 | I think about my rosacea |
| 21 | I avoid certain environments (heat, humidity, cold) because of my rosacea |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.6.3.2: RosaQoL (Page xx of yy)

| S: Subject | | SGT-54-07 | Data of | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| A: Age/Sex<br>E: Eval | Visit | Analysis Visit | Date of | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 1 2 | 1 2 | 1 / | 15 | 16 | 17 | 10 | 1 0 | 20 | 21 |
| | VISIC | Analysis visit | Assessment | 1 | | | | | | | | | | | 12 | 13 | 14 | 1.0 | 10 | | 10 | | | |
| S: xxxxxx | xxxxxxx | xxxxxxxxx | xxxxxxxxx | Х | Х | Х | Х | Х | Х | Х | х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| A: xxx | | | | | | | | | | | | | | | | | | | | | | | | |
| E: x | | | | | | | | | | | | | | | | | | | | | | | | |
| | XXXXXXX | XXXXXXXXX | XXXXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | XXXXXXX | XXXXXXXXX | XXXXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | Х | Х | Х | Х | X | Х | Х | Х | X | Х |
| | XXXXXXXX | XXXXXXXXX | XXXXXXXXX | Х | Х | Х | Х | Х | Х | X | X | X | X | X | X | Х | X | Х | X | Х | Х | Х | X | Х |
| | XXXXXXXX | XXXXXXXXX | XXXXXXXXX | Х | X | X | Х | Х | Х | X | X | X | X | Х | X | X | X | X | X | X | X | Х | X | Х |
| | XXXXXXXX | XXXXXXXXX | XXXXXXXXX | Х | X | X | Х | Х | Х | X | X | X | X | Х | X | X | X | X | X | X | X | Х | X | Х |
| | XXXXXXXX | XXXXXXXXX | XXXXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | Х | Х | Х | Х | Х |
| S: xxxxxx | XXXXXXX | xxxxxxxxx | xxxxxxxxx | Х | Х | Х | х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х | Х | Х | Х | Х | х |
| A: xxx | | | | | | | | | | | | | | | | | | | | | | | | |
| E: x | | | | | | | | | | | | | | | | | | | | | | | | |
| | XXXXXXXX | XXXXXXXXX | XXXXXXXXX | Х | X | X | Х | Х | Х | X | X | X | X | X | X | Х | X | X | X | Х | X | Х | Х | Х |
| | XXXXXXXX | XXXXXXXXX | XXXXXXXXX | X | X | X | X | Х | Х | X | X | X | X | X | X | X | X | X | X | X | X | Х | X | Х |
| | XXXXXXXX | XXXXXXXXX | XXXXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | X | X | Х | Х | Х | Х | Х | X | Х | Х | Х | X | Х |
| | XXXXXXXX | XXXXXXXXX | XXXXXXXXX | Х | X | X | Х | Х | Х | X | X | X | X | X | X | Х | X | X | X | Х | X | Х | Х | Х |
| | XXXXXXXX | XXXXXXXXX | XXXXXXXXX | X | X | X | X | Х | Х | X | X | X | X | X | X | X | X | X | X | X | X | Х | X | Х |
| | XXXXXXXX | xxxxxxxxx | xxxxxxxxx | X | X | X | X | Х | Х | Х | Х | Х | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| S: xxxxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | х | х | х | х | Х | Х | х | Х | Х | Х | Х | Х | х | Х | Х | Х | Х | Х | Х | х | х |
| A: xxx<br>E: x | | | | | | | | | | | | | | | | | | | | | | | | |
| | xxxxxxx | xxxxxxxxx | xxxxxxxxx | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х |
| | XXXXXXX | XXXXXXXXX | xxxxxxxxx | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | XXXXXXX | XXXXXXXXX | XXXXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | XXXXXXX | XXXXXXXXX | XXXXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | XXXXXXX | XXXXXXXXX | XXXXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | XXXXXXXX | xxxxxxxxx | XXXXXXXXX | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| A: xxx | ********* ********* ******** | ************************************** | ************************************** | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | x<br>x<br>x<br>x | X<br>X<br>X<br>X | X<br>X<br>X<br>X | X<br>X<br>X<br>X | х<br>х<br>х<br>х | |

 $<sup>\</sup>overline{1}$  = Never; 2 = Rarely; 3 = Sometimes; 4 = Often; 5 = All the time; ND = Not Done Note: Full RosaQoL question text is available in Listing 16.2.6.3.1.

### Listing sorted by Subject and Visit Number

Listing 16.2.6.3.3: RosaQoL Subscales Scores (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | SGT-54-07<br>Analysis Visit | Date of<br>Assessment | Total Score <sup>1</sup> | Symptom <sup>2</sup> | Functional <sup>3</sup> | Emotional <sup>4</sup> |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxx | xxxxxxxx | xxxxxxxx | x xxxxxxxxx | xxxxxxxxx | xx | xx | xx | xx |
| | | | xxxxxxxx | x xxxxxxxxx | xxxxxxxxx | XX | XX | xx | XX |
| | | | xxxxxxxx | x xxxxxxxxx | XXXXXXXXX | XX | XX | xx | XX |
| | | | xxxxxxxx | x xxxxxxxxx | xxxxxxxxx | xx | xx | XX | xx |
| xxxxxx | xxxxx | xxxxxxx | xxxxxxxx | x xxxxxxxxx | xxxxxxxxx | xx | xx | XX | xx |
| | | | XXXXXXXX | x xxxxxxxxx | XXXXXXXXX | XX | XX | XX | XX |
| | | | XXXXXXXX | X XXXXXXXXX | XXXXXXXXX | XX | XX | XX | XX |
| | | | XXXXXXXX | x xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| xxxxxx | XXXXX | xxxxxxx | xxxxxxxx | x xxxxxxxxx | xxxxxxxxx | xx | xx | xx | xx |
| | | | XXXXXXXX | x xxxxxxxxx | XXXXXXXXX | XX | XX | XX | XX |
| | | | XXXXXXXX | X XXXXXXXXX | XXXXXXXXX | XX | XX | XX | XX |
| | | | XXXXXXXX | x xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| xxxxxx | XXXXX | xxxxxxx | xxxxxxxx | x xxxxxxxxx | xxxxxxxxx | xx | xx | xx | xx |
| | | | XXXXXXXX | x xxxxxxxxx | XXXXXXXXX | XX | XX | xx | XX |
| | | | XXXXXXXX | x xxxxxxxxx | XXXXXXXXX | XX | XX | xx | XX |
| | | | xxxxxxxx | x xxxxxxxxx | xxxxxxxxx | xx | xx | XX | XX |
| xxxxxx | xxxxx | xxxxxxx | xxxxxxxx | x xxxxxxxxx | xxxxxxxxx | xx | xx | XX | xx |
| | | | xxxxxxxx | x xxxxxxxx | XXXXXXXXX | XX | XX | XX | XX |
| | | | xxxxxxxx | x xxxxxxxxx | XXXXXXXXX | XX | XX | XX | XX |
| | | | XXXXXXXX | x xxxxxxxxx | XXXXXXXXX | XX | XX | XX | XX |

Total Score calculated from the unweighted mean of all RosaQoL questions.

#### Listing sorted by Subject and Visit Number

<sup>&</sup>lt;sup>2</sup> Symptom Subscale Score calculated from items 2, 6, 9, 16, 17, 18, and 19. <sup>3</sup> Functional Subscale Score calculated from items 13, 15, and 21.

 $<sup>^4</sup>$  Emotional Subscale Score calculated from items 1, 3, 4, 5, 7, 8, 10, 11, 12, 14, and 20.

Listing 16.2.6.4: Erythema Severity/Telangiectasia Assessments (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | SGT-54-07<br>Analysis Visit | Date of<br>Assessment | Evaluator<br>Initials | Assessment | Result |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxx | xxx | Rosacea Erythema<br>Telangiectasia | ********* |
| | | | XXXX X | xxxx x | xxxxxxxxx | xxx | Rosacea Erythema<br>Telangiectasia | xxxxxxxxx |
| | | | XXXX X | xxxx x | xxxxxxxxx | xxx | Rosacea Erythema<br>Telangiectasia | xxxxxxxxx<br>xxxxxxxx |
| | | | XXXX X | xxxx x | xxxxxxxxx | xxx | Rosacea Erythema<br>Telangiectasia | xxxxxxxxx |
| | | | xxxx x | xxxx x | xxxxxxxxx | xxx | Rosacea Erythema<br>Telangiectasia | xxxxxxxxx<br>xxxxxxxx |
| | | | xxxx x | xxxx x | xxxxxxxxx | xxx | Rosacea Erythema<br>Telangiectasia | xxxxxxxxx |
| | | | XXXX X | xxxx x | xxxxxxxxx | xxx | Rosacea Erythema<br>Telangiectasia | ******** |

Listing sorted by Subject and Visit Number, and Assessment (in order presented on eCRF).

Listing 16.2.7.1: Cutaneous Safety and Tolerability Assessments (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | SGT-54-07<br>Analysis Visit | Date of<br>Assessment | Evaluator<br>Initials | Test | Result |
|---|---|---|---|---|---|---|---|---|
| XXXXX | xxxx | xxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | XXX | Dryness | xxxxxxx |
| | | | | | | | Scaling | xxx xxxx |
| | | | | | | | Itching | xxxxxxxxxxx |
| | | | | | | | Burning/Stinging | xxxxxxxxxx |
| | | | xxxx x | xxxx x | xxxxxxxxx | xxx | Dryness | xxxxxxx |
| | | | | | | | Scaling | xxx xxxx |
| | | | | | | | Itching | xxxxxxxxxx |
| | | | | | | Burning/Stinging | xxxxxxxxx | |
| | | | xxxx x | xxxx x | xxxxxxxxx | xxx | Dryness | xxxxxxx |
| | | | | | | | Scaling | xxx xxxx |
| | | | | | | | Itching | XXXXXXXXX |
| | | | | | | | Burning/Stinging | XXXXXXXXXX |
| | | | xxxx x | xxxx x | xxxxxxxxx | xxx | Dryness | xxxxxxx |
| | | | | | | | Scaling | xxx xxxx |
| | | | | | | | Itching | xxxxxxxxxx |
| | | | | | | | Burning/Stinging | XXXXXXXXXX |
| | | | xxxx x | XXXX X | xxxxxxxxx | XXX | Dryness | XXXXXXX |
| | | | | | | | Scaling | XXX XXXX |
| | | | | | | | Itching | XXXXXXXXXX |
| | | | | | | | Burning/Stinging | XXXXXXXXXX |
| | | | XXXX X | XXXX X | XXXXXXXXX | XXX | Dryness | XXXXXXX |
| | | | | | | | Scaling | XXX XXXX |
| | | | | | | | Itching | XXXXXXXXXX |
| | | | | | | | Burning/Stinging | xxxxxxxxx |

Listing sorted by Subject, Visit Number, and Test (in order presented on eCRF).

Listing 16.2.7.2.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Application<br>Area | Adverse Event |
|---|---|---|---|
| ******* | ******** | xxx | ********** |
| | | xx | xxxxxxxx |
| | | xx | xxxxx xxxxxxxx |
| | xxxxxxxx | xx | xxxxxxx |
| ***** | xxxxxxx | xx | xxxxxxx |
| *** *** ********* | xxxxxx | xxx | xxxxxxxx xx xxxxxxx |
| | xxxx xxxxxxxxxx | xx | xxxxxx xxxx xxxxxxxx xxx |


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by System Organ Class, Preferred Term, Adverse Event.

### Listing 16.2.7.2.2: Pre-Treatment Adverse Events (Page xx of yy)

| S: Subject<br>A: Age/Sex | S: MedDRA System Organ Class<br>P: MedDRA Preferred Term | A: In the Application Area G: Severity R: Relationship to Study Drug | Τ: | | S: | |
|---|---|---|---|---|---|---|
| E: Eval | A: Adverse Event | S: Serious Event | 0: | Outcome | E: | End Date (Day) 1 |
| S: xxxxxx | S: xxxx xxx xxxxxxxxxx xxxxx | A: xx | A: | xxx xx xxxxxxx | s: | xxxxxxxxxxxx |
| A: xxxx | P: xxx xxxxxxxxxx | G: xxxx | Т: | xxxx | E: | xxxxxxxxxxxxx |
| E: xxxxxxxx | A: xxxxxxx xxxx xxxxxxxx xxxxx | R: xxx xxxxxxx<br>S: xx | 0: | xxxxxxxxxxxxxx | | |
| | S: xxxxxx xxxxxxxx xxx xxxxxxxx | A: xxx | A: | xxx xxxxxxxxx | S: | xxxxxxxxxxxx |
| | P: xxxxxxxxx | G: xxxx | Т: | xxxxxxxxxx xxxxxxxx | E: | xxxxxxxxxxxxx |
| | A: xxxxxxx xxxxx xxxxx xxxx | R: xxx xxxxxxx<br>S: xx | 0: | xxxxxxxxxxxxxx | | |
| S: xxxxxx | S: xxxx xxxxxxxx xxxxx | A: xx | A: | xxx xx xxxxxxx | s: | xxxxxxxxxxxx |
| A: xxxx | P: xxxxxxxx | G: xxxxxxxx | Т: | XXXX | E: | xxxxxxxxxxxx |
| E: xxxxxxx | A: xxxxxxxx xxxxx | R: xxx xxxxxxx<br>S: xx | 0: | xxxxxxxxxxxxxx | | |
| S: xxxxxx | S: xxxx xxxxxxxx xxxxx | A: xx | A: | xxx xx xxxxxxx | s: | xxxxxxxxxxxx |
| A: xxxx | P: xxxxxxxx | G: xxxxxxxx | Т: | XXXX | E: | XXXXXXXXXXXXX |
| E: xxxxxxx | A: xxxxxxxx xxxxx | R: xxxxxxx<br>S: xxx | 0: | xxxxxxxxxxxxxx | | |
| | S: xxxxxx xxxxxxx xxx xxxxxxxx | A: xxx | A: | xxx xxxxxxxxx | S: | xxxxxxxxxxxx |
| | P: xxxxxxxxx | G: xxxx | Τ: | XXXXXXXXXX XXXXXXXX | E: | XXXXXXXXXXXXX |
| | A: xxxxxxx xxxxx xxxxxx xxxx | R: xxx xxxxxxx<br>S: xx | 0: | xxxxxxxxxxxxxx | | |

<sup>1</sup> Day is calculated as date - date of first application of E-BPO 5% Cream (from SGT-54-01/SGT-54-02 or SGT-54-07) for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

### Listing 16.2.7.2.3: Treatment-Emergent Adverse Events (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | S: MedDRA System Organ Class P: MedDRA Preferred Term A: Adverse Event | A: In the Application Area G: Severity R: Relationship to Study Dru S: Serious Event | A: Action Taken with Study Drug T: Action Taken to Treat Event O: Outcome | |
|---|---|---|---|---|
| S: xxxxx | S: xxxx xxx xxxxxxxxxx xxxxx | A: xx | A: xxx xx xxxxxxx | S: xxxxxxxxxxxxx |
| A: xxxx<br>E: xxxxxxx | P: xxx xxxxxxxxxxx<br>A: xxxxxxx xxxx xxxxxxxx xxxxx | G: xxxx<br>R: xxx xxxxxxx<br>S: xx | T: xxxx<br>O: xxxxxxxxxxxxxxxxxx | E: xxxxxxxxxxxxxxx |
| | S: xxxxxxx xxxxxxxx xxx xxxxxxxx<br>P: xxxxxxxxx<br>A: xxxxxxxx xxxx xxxxx xxxxxx | A: xxx<br>G: xxxx<br>R: xxx xxxxxxx<br>S: xx | A: xxx xxxxxxxxxx<br>T: xxxxxxxxxxx xxxxxxxx<br>O: xxxxxxxxxxxxxx | S: xxxxxxxxxxxxxxx<br>E: xxxxxxxxxxxxxxxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | S: xxxx xxxxxxxx xxxxxx P: xxxxxxxxx A: xxxxxxxx xxxxx | A: xx<br>G: xxxxxxxx<br>R: xxx xxxxxxx<br>S: xxx | A: xxx xx xxxxxxx<br>T: xxxx<br>O: xxxxxxxxxxxxxxxxx | S: xxxxxxxxxxxxxxx<br>E: xxxxxxxxxxxxxxxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | S: xxxx xxxxxxxx xxxxxx<br>P: xxxxxxxxx<br>A: xxxxxxxx xxxxx | A: xx<br>G: xxxxxxxx<br>R: xxx xxxxxxx<br>S: xxx | A: xxx xx xxxxxxx<br>T: xxxx<br>O: xxxxxxxxxxxxxxxxx | S: xxxxxxxxxxxxxxx<br>E: xxxxxxxxxxxxxxxxx |
| | S: xxxxxxx xxxxxxxx xxx xxxxxxxx<br>P: xxxxxxxxx<br>A: xxxxxxxx xxxx xxxxx xxxxx | A: xxx<br>G: xxxx<br>R: xxxxxxx<br>S: xx | A: xxx xxxxxxxxxx<br>T: xxxxxxxxxxx xxxxxxxx<br>O: xxxxxxxxxxxxxx | S: xxxxxxxxxxxxxxxx<br>E: xxxxxxxxxxxxxxxxxx |

Day is calculated as date - date of first application of E-BPO 5% Cream (from SGT-54-01/SGT-54-02 or SGT-54-07) for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

### Listing 16.2.7.2.4: Serious Adverse Events (Page xx of yy)

| S: Subject | S: MedDRA System Organ Class P: MedDRA Preferred Term A: Adverse Event | A: In the Application Area<br>G: Severity | A: Action Taken with Study Druc | ı |
|---|---|---|---|---|
| A: Age/Sex | O: Occurred Prior to First | R: Relationship to Study Drug | T: Action Taken to Treat Event | S: Start Date (Day) 1 |
| E: Eval | Application | S: Serious Event | O: Outcome | E: End Date (Day) 1 |
| S: xxxxxx | S: xxxx xxx xxxxxxxxxx xxxxx | A: xx | A: xxx xx xxxxxxx | S: xxxxxxxxxxxxx |
| A: xxxx | P: xxx xxxxxxxxxx | G: xxxx | T: xxxx | E: xxxxxxxxxxxxxx |
| E: xxxxxxxx | A: xxxxxxx xxxx xxxxxxxx xxxxx | R: xxx xxxxxxx | O: xxxxxxxxxxxxxxx | |
| | 0: xx | S: xxx | | |
| | S: xxxxxx xxxxxxx xxx xxxxxxxx | A: xxx | A: xxx xxxxxxxxx | S: xxxxxxxxxxxxxx |
| | P: xxxxxxxxx | G: xxxx | T: xxxxxxxxxx xxxxxxxx | E: xxxxxxxxxxxxxx |
| | A: xxxxxxxx xxxxx xxxxxx xxxx | R: xxx xxxxxxx | O: xxxxxxxxxxxxxxxx | |
| | 0: xx | S: xxx | | |
| S: xxxxxx | S: xxxx xxxxxxxx xxxxx | A: xx | A: xxx xx xxxxxxx | S: xxxxxxxxxxxxxx |
| A: xxxx | P: xxxxxxxx | G: xxxxxxxx | T: xxxx | E: xxxxxxxxxxxxxx |
| E: xxxxxxxx | A: xxxxxxxx xxxxx | R: xxxxxxx | O: xxxxxxxxxxxxxxxx | |
| | O: xx | S: xxx | | |


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

<sup>1</sup> Day is calculated as date - date of first application of E-BPO 5% Cream (from SGT-54-01/SGT-54-02 or SGT-54-07) for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.

Listing 16.2.7.2.5: Subjects Who Prematurely Discontinued Study and/or Discontinued Study Drug Due to Adverse Events (Page xx of yy)

| S: Subject | S: MedDRA System Organ Class P: MedDRA Preferred Term A: Adverse Event | A: In the Application Area<br>G: Severity | A: Action Taken with Study Drug | ı |
|---|---|---|---|---|
| A: Age/Sex<br>E: Eval | O: Occurred Prior to First Application | R: Relationship to Study Drug<br>S: Serious Event | T: Action Taken to Treat Event O: Outcome | S: Start Date (Day) <sup>1</sup><br>E: End Date (Day) <sup>1</sup> |
| S: xxxxx | S: xxxx xxx xxxxxxxxx xxxxx | A: xx | A: xxx xx xxxxxxx | S: xxxxxxxxxxxx |
| A: xxxx | P: xxx xxxxxxxxxx | G: xxxx | T: XXXX | E: XXXXXXXXXXXXXXX |
| E: xxxxxxxx | A: xxxxxx xxxx xxxxxxx xxxx | R: xxx xxxxxxx | 0: xxxxxxxxxxxxxx | <b>.</b> |
| _, | 0: xx | S: xxx | | |
| | S: xxxxxx xxxxxxx xxx xxxxxxx | A: xxx | A: xxx xxxxxxxxx | S: xxxxxxxxxxxxxx |
| | P: xxxxxxxxx | G: xxxx | T: xxxxxxxxxx xxxxxxxx | E: xxxxxxxxxxxxxx |
| | A: xxxxxxxx xxxxx xxxxxx xxxx | R: xxx xxxxxxx | O: xxxxxxxxxxxxxxxx | |
| | O: xx | S: xxx | | |
| S: xxxxxx | S: xxxx xxxxxxxx xxxxx | A: xx | A: xxx xx xxxxxxx | S: xxxxxxxxxxxxxx |
| A: xxxx | P: xxxxxxxx | G: xxxxxxxx | T: xxxx | E: xxxxxxxxxxxxxx |
| E: xxxxxxxx | A: xxxxxxxx xxxxx | R: xxxxxxx | O: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | |
| | O: xx | S: xxx | | |


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

<sup>1</sup> Day is calculated as date - date of first application of E-BPO 5% Cream (from SGT-54-01/SGT-54-02 or SGT-54-07) for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.

Listing 16.2.8.1: Urine Pregnancy Tests (Page xx of yy)

| ubject | Age/Sex | Eval | Visit | Date of Assessment | Results | Reason Test Not Done |
|---|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | xxxxxxx | |
| | | | xxxxxxxx | xxxxxxxxx | XXXXXXXX | |
| | | | xxxx x | | | xxx xxxx |
| | | | xxxx x | xxxxxxxxx | XXXXXXXX | |
| | | | XXXX XX | xxxxxxxxx | XXXXXXX | |
| | | | XXXX XX | xxxxxxxxx | XXXXXXX | |
| | | | xxxx xx | xxxxxxxxx | XXXXXXXX | |
| | | | XXXX XX | xxxxxxxxx | XXXXXXX | |
| | | | xxxx xx | xxxxxxxxx | XXXXXXX | |
| | | | xxxx xx | xxxxxxxxx | XXXXXXX | |
| | | | XXXX XX | xxxxxxxxx | xxxxxxx | |
| ΧX | XXXX | xxxxxxx | xxxxxxxx | xxxxxxxxx | xxxxxxx | |
| | | | xxxxxxx | xxxxxxxxx | XXXXXXX | |
| | | | XXXX X | XXXXXXXXX | XXXXXXX | |
| | | | XXXX X | XXXXXXXXX | XXXXXXX | |
| | | | XXXX XX | XXXXXXXXX | XXXXXXX | |
| | | | XXXX XX | XXXXXXXXX | XXXXXXX | |
| | | | XXXX XX | XXXXXXXXX | XXXXXXX | |
| | | | XXXX XX | XXXXXXXXX | XXXXXXXX | |
| | | | XXXX XX | XXXXXXXXX | XXXXXXXX | |
| | | | XXXX XX | XXXXXXXXX | XXXXXXXX | |
| | | | XXXX XX | xxxxxxxxx | XXXXXXX | |
| XΧ | XXXX | xxxxxxx | xxxxxxxx | | | xxx xxxxxxxxx |
| | | | xxxxxxxx | | | XXX XXXXXXXXX |
| | | | XXXX X | | | XXX XXXXXXXXX |
| | | | xxxx x | | | XXX XXXXXXXXX |
| | | | XXXX XX | | | XXX XXXXXXXXX |
| | | | xxxx xx | xxxxxxxxx | XXXXXXXX | |
| | | | xxxx xx | xxxxxxxx | XXXXXXX | |
| | | | xxxx xx | xxxxxxxxx | XXXXXXX | |
| | | | xxxx xx | xxxxxxxxx | XXXXXXX | |
| | | | xxxx xx | xxxxxxxxx | XXXXXXX | |
| | | | XXXX XX | XXXXXXXXX | XXXXXXX | |

Listing sorted by Subject and Visit Number.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

# Listing 16.2.8.2: Physical Examination (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of<br>Assessment | Body System | Exam Finding | Reason Exam<br>Not Done |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxx | xxxxxxxxx | xxxxx<br>xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXX<br>XXXXXX<br>XXXXXXX XXXXXXXXX XXXX<br>XXXXXX XXXXX XXXX XXXX | |
| | | | xxxx xxxxx | xxxxxxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxx xxxx<br>xxx xxxx<br>xxx xxxx | xxx xxxxxxxxx<br>xxx xxxxxxxxx |
| xxxxx | xxxxx xxxx | xxxxxxx | xxxxxxx | xxxxxxxxx | xxxxx<br>xxxxxx<br>xxxxxxx<br>xxxxxxxxxxxxxxxxx | ****** ****** ****** ****** ****** **** | |
| | | | xxxx xxxxx | xxxxxxxxx | xxxx<br>xxxxxxxxxxxx<br>xxxxxxxxxxxx<br>xxxxxxxx | xxx xxxx<br>xxx xxxx<br>xxx xxxx | xxx xxxxxxxxx<br>xxx xxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit Number, and Body System (in order presented on eCRF).

Listing 16.2.8.3: Vital Signs (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of<br>Assessment | Vital Sign | Result | Units |
|---|---|---|---|---|---|---|---|
| XXXXXX | xxxx | xxxxxxx | xxxxxxx | xxxxxxxxx | ****** | xx | xxxx |
| | | | | *************************************** | XXXXX XXXX | XX | XXXXXXXXX |
| | | | | | xxxxxx | xxxxx | XX |
| | | | | | xxxxxxxxxx xxxx | XX | XXXXXXXXXX |
| | | | | | xxxxxxx xxxxx xxxxxxx | XXX | XXXX |
| | | | | | xxxxxxxxxx | XXXX | Х |
| | | | | | xxxxxx | xxx | XX |
| | | | xxxx xxxxx | xxxxxxxxx | ****** | xx | xxxx |
| | | | | | XXXXX XXXX | XXX XXXX | |
| | | | | | xxxxxxxxxx xxxx | xxx | XXXXXXXXXX |
| | | | | | xxxxxxx xxxxx xxxxxxx | xxx | XXXX |
| | | | | | xxxxxxxxx | xx | Х |
| XXXXX | xxxx | xxxxxxx | xxxxxxx | xxxxxxxxx | xxxxxxxx xxxxx xxxxxxx | xx | xxxx |
| | | | | | XXXXX XXXX | XX | XXXXXXXX |
| | | | | | XXXXXX | XXX | XX |
| | | | | | xxxxxxxxxx xxxx | XX | XXXXXXXXXX |
| | | | | | xxxxxxx xxxxx xxxxxxx | XX | XXXX |
| | | | | | XXXXXXXXX | XX | X |
| | | | | | xxxxxx | xxx | XX |
| | | | xxxx xxxxx | xxxxxxxxx | xxxxxxxx xxxxx xxxxxxx | xxx xxxx | |
| | | | | | XXXXX XXXX | XXX XXXX | |
| | | | | | XXXXXXXXXX XXXX | XXX XXXX | |
| | | | | | XXXXXXX XXXXX XXXXXXX | XXX XXXX | |
| | | | | | XXXXXXXXX | XXX XXXX | |

Listing sorted by Subject, Visit Number, and Vital Sign (in alphabetical order).